CLINICAL TRIAL: NCT01393639
Title: A PHASE 2, RANDOMIZED, DOUBLE BLIND ASSESSMENT OF EFFICACY AND SAFETY OF PF 04171327(1, 5, 10, 15 MG DOSE, DAILY) COMPARED TO 5 MG AND 10 MG PREDNISONE DAILY AND PLACEBO DAILY IN SUBJECTS WITH RHEUMATOID ARTHRITIS OVER AN 8 WEEK PERIOD FOLLOWED BY A 4 WEEK PERIOD OF TAPERING OF STUDY DRUG.
Brief Title: Study Comparing Doses Of An Experimental Glucocorticoid Compound To Prednisone And Placebo In Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A9391010; 2010-023782-22 (EudraCT Number)
Record Dates: First submitted 2011-06-13; First posted 2011-07-13 (Estimated); Results first posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Rheumatoid Arthritis
Keywords: treatment of rheumatoid arthritis; treatment of RA; patients on methotrexate for rheumatoid arthritis; prednisone for rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — fosdagrocorat; Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- PF-04171327 1 mg QD (Experimental)
  Interventions: Drug: PF-04171327
- PF-04171327 5 mg QD (Experimental)
  Interventions: Drug: PF-04171327
- PF-04171327 10 mg QD (Experimental)
  Interventions: Drug: PF-04171327
- PF-04171327 15 mg QD (Experimental)
  Interventions: Drug: PF-04171327
- prednisone 5 mg QD (Active Comparator)
  Interventions: Drug: prednisone
- prednisone 10 mg QD (Active Comparator)
  Interventions: Other: prednisone
- placebo (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: PF-04171327 — 1 mg tablet once daily (QD) for 8 weeks
  Arms: PF-04171327 1 mg QD
Drug: PF-04171327 — 5 mg tablet once daily (QD) for 8 weeks
  Arms: PF-04171327 5 mg QD
Drug: PF-04171327 — 10 mg tablet once daily (QD) for 8 weeks
  Arms: PF-04171327 10 mg QD
Drug: PF-04171327 — 15 mg tablet once daily (QD) for 8 weeks
  Arms: PF-04171327 15 mg QD
Drug: prednisone — 5 mg capsule once daily for 8 weeks
  Arms: prednisone 5 mg QD
Other: prednisone — 10 mg capsule once daily for 8 weeks
  Arms: prednisone 10 mg QD
Other: placebo — placebo (tablet or capsule) once daily (QD) for 8 weeks
  Arms: placebo

SUMMARY:
The purpose of this study is to compare the safety and efficacy of multiple doses of PF-04171327, an experimental glucocorticoid drug, to prednisone at 5 mg or 10 mg and placebo in the treatment of rheumatoid arthritis. All subjects will also be receiving background treatment of methotrexate for their rheumatoid arthritis. Study medication will be given for eight weeks followed by a 4 week period during which the dose of study medication will be gradually reduced. The efficacy of the study medications will be determined by assessing severity of the rheumatoid arthritis during the study and safety will be determined by adverse event reporting, laboratory tests and biomarker analysis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have documented rheumatoid arthritis with a duration of at least 3 months as determined by the investigator using standardly accepted criteria, must have been receiving methotrexate for at least 3 months to treat their rheumatoid arthritis, and must be free of any signs or symptoms of infection.

Exclusion Criteria:

* Subjects cannot enter the study if they have recently received treatment with certain medications which might interfere with study medications;
* subjects cannot enter if they have abnormalities in certain blood tests, history of cancer, recent bone fracture or other significant conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2011-09-27 (Actual); Primary Completion 2014-06-03 (Actual); Study Completion 2014-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (93):
- United States (14):
  - Catalina Pointe Clinical Research, Inc., Tucson, Arizona
  - C. Michael Neuwelt, MD, Inc., San Leandro, California
  - Javed Rheumatology Associates, Inc., Newark, Delaware
  - Allergy, Asthma, Arthritis, and Lung Center, Daytona Beach, Florida
  - Millennium Research, Ormond Beach, Florida
  - Alastair C. Kennedy, MD, Vero Beach, Florida
  - The Center for Arthritis and Rheumatism, Vero Beach, Florida
  - Arthritis and Osteoporosis Medical Associates, PLLC, Brooklyn, New York
  - Cincinnati Rheumatic Disease Study Group, Inc., Cincinnati, Ohio
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Low Country Rheumatology, PA, Charleston, South Carolina
  - Tricounty Radiology, Charleston, South Carolina
  - Accurate Clinical Research, Inc., Houston, Texas
  - Arthritis Northwest, PLLC, Spokane, Washington
- Bulgaria (4):
  - Revmatologichen kabinet, DKTs Sv. Pantaleimon OOD, Pleven
  - Revmatologichno Otdelenie, MBAL - Plovdiv, Plovdiv
  - MBAL "Sveti Ivan Rilski" Sofia; Klinika po Revmatologia, Sofia
  - MBAL Sveti Ivan Rilski Sofia; Klinika po Revmatologia, Sofia
- Colombia (4):
  - Hospital Pablo Tobon Uribe, Medellín, Antioquia
  - Reumalab S.A.S, Medellín, Antioquia
  - Centro Integral de Reumatologia e Inmunologia CIREI, Bogota, Cundinamarca
  - Preventive Care SAS, Chía, Cundinamarca
- Czechia (4):
  - Revmatologie Bruntal, S.R.O., Bruntál
  - Revmatologicka ambulance, Ostrava - Poruba
  - Revmatologicka ambulance, Prague
  - Thomayerova nemocnice, Prague
- Germany (3):
  - Charite Universitaetsmedizin Berlin, Klinik fuer Rheumatologie, Berlin
  - Klinische Forschung Berlin-Buch GmbH, Berlin
  - CIRI GmbH, Frankfurt am Main
- Hungary (6):
  - Dr. Rethy Pal Korhaz es Rendelointezet, II. Reumatologia Szakrendeles, Békéscsaba
  - Budai Irgalmasrendi Korhaz, Reumatologia I., Budapest
  - Revita Reumatologiai Rendelo, Budapest
  - Qualiclinic Kft., Budapest
  - Fejer Megyei Szent Gyorgy Korhaz Reumatologia, Székesfehérvár
  - MAV Korhaz es Rendelointezet, Reumatologiai szakrendeles, Szolnok
- India (3):
  - Krishna Institute of Medical Sciences Ltd, Secunderabad, Andhra Pradesh
  - Shirdi Sai Hospital, Bangalore, Karnataka
  - Dapartment of Rheumatology, Lucknow, Uttar Pradesh
- Malaysia (2):
  - Hospital Raja Permaisuri Bainun, Ipoh, Perak
  - Sunway Medical Centre, Petaling Jaya, Selangor
- Mexico (3):
  - Centro de Estudios de Investigacion Basica y Clinica SC., Guadalajara, Jalisco
  - Unidad de Investigacion Biomedica del CEM, Mérida, Yucatán
  - Centro de Alta Especialidad en Reumatologia e Investigacion del Potosi S.C., San Luis Potosí City
- Poland (3):
  - Centrum Kliniczno-Badawcze J. Brzezicki, B. Górniakiewicz-Brzezicka Lekarze Spółka Partnerska, Elblag
  - Nzoz "Lecznica Mak-Med S.C.", Nadarzyn
  - Wojewodzki Zespol Reumatologiczny im. dr J. Titz-Kosko, Sopot
- Romania (4):
  - Spitalul Clinic "Sfanta Maria", Clinica de Medicina Interna si Reumatologie, Bucharest
  - Spitalul Clinic Judetean de Urgenta "Sfantul Apostol Andrei", Galati
  - Spitalul Clinic de Recuperare, Iași
  - Spitalul Clinic Judetean de Urgenta Targu Mures, Reumatologic, Tg Mures
- Russia (18):
  - GBOU VPO "Orenburg State Medical Academy of Ministry of Healthcare of Russian Federation", Orenburg, Russian Federation
  - Territorial Clinical Hospital, Barnaul
  - GBUZ of Kemerovo region Regional clinical hospital for was veterans, Kemerovo
  - Kemerovo Regional Clinical Hospital, Kemerovo
  - FSBI Scientific - Research Institute of Rheumatology RAMS n.a. V.A. Nasonova., Moscow
  - LLC Consultative and Diagnostic Rheumatological Center Healthy Joints, Novosibirsk
  - Republican Hospital V.A.Baranov, Petrozavodsk
  - Ryazan Regional Clinical Cardiological Dispensary, Ryazan
  - Clinical Rheumatological Hospital #25, Saint Petersburg
  - Clinical Hospital #122 L.G. Sokolov, Saint Petersburg
  - MUZ City Clinical Hospital #12, Saratov
  - Smolensk Regional Clinical Hospital, Smolensk
  - Tomsk Regional Clinical Hospital, Tomsk
  - Vladimir Regional Clinical Hospital, Vladimir
  - Clinical Hospital of Emergency Care N.V. Soloviev, Yaroslavl
  - Yaroslavl Regional Clinical Hospital, Yaroslavl
  - Sverdlovsk Regional Clinical Hospital # 1, Yekaterinburg
  - Municilap Institution Central Clinical Hospital 6, Yekaterinburg
- Serbia (2):
  - Institute of Rheumatology, Belgrade
  - Institute for treatment and rehabilitation Niska Banja, Niška Banja
- Slovakia (5):
  - AAGS, s.r.o. , nestatne zdravotnicke zariadenie, Dunajská Streda
  - Nestatna reumatologicka ambulancia, Považská Bystrica
  - Reumatologicka ambulancia, REUMEX, s.r.o., Rimavská Sobota
  - Reumaglobal s.r.o., Trnava
  - Nestatna reumatologicka ambulancia, Žilina
- South Africa (2):
  - Panorama Medical Centre, Panorama, Cape Town
  - Emmed Research, Pretoria, Gauteng
- South Korea (5):
  - KyungHee University Hospital, Seoul, Korea
  - Daegu Catholic University Medical Center, Department of Rheumatology, Daegu
  - Inha University Hospital, Medicine/Rheumatology, Incheon
  - Seoul National University Hospital, Rheumatology, Internal Medicine, Seoul
  - Konkuk University Medical Center, Department of Rheumatology, Seoul
- Spain (2):
  - Complejo Hospitalario Universitario A Coruña. Hospital Materno Infantil Teresa Herrera, A Coruña
  - Hospital SANITAS CIMA., Barcelona
- Ukraine (9):
  - Municipal Medical Institution "City Clinical Hospital #3", Chernivtsi
  - Municipal Medicoprophylactic Institution "Donetsk City Clinical Hospital #5"., Donetsk
  - National Scientific Centre "Institute of Cardiology n.a. M.D. Strazheska of NAMS of Ukraine"., Kiev
  - Komunalnyi zaklad Kyivskoi oblasnoi rady "Kyivska oblasna klinichna likarnia", Kyiv
  - Komunalnyi zaklad Lvivskoi oblasnoi rady "Lvivskyi oblasnyi klinichnyi diahnostychnyi tsentr", Lviv
  - Komunalna ustanova "Odeska oblasna klinichna likarnia", Odesa
  - Municipal Establishment "City Clinical Hospital #9 n.a. O.I. Minakov", Department of Rheumatology, Odesa
  - Vinnytsya regional clinical hospital named after M.I. Pyrogova; Department of rheumatology, Vinnytsia
  - Municipal Institution:"Zaporizhzhya Regional Clinical Hospital",Rheumatology Dep., Zaporizhzhya

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Buttgereit F, Strand V, Lee EB, Simon-Campos A, McCabe D, Genet A, Tammara B, Rojo R, Hey-Hadavi J. Fosdagrocorat (PF-04171327) versus prednisone or placebo in rheumatoid arthritis: a randomised, double-blind, multicentre, phase IIb study. RMD Open. 2019 Apr 16;5(1):e000889. doi: 10.1136/rmdopen-2018-000889. eCollection 2019. PMID 31168411
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9391010&StudyName=Study%20Comparing%20Doses%20Of%20An%20Experimental%20Glucocorticoid%20Compound%20To%20Prednisone%20And%20Placebo%20In%20Rheumatoid%20Arthritis%20

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multi-center, randomized, double-blind, parallel-group, active and placebo-controlled study randomized 323 participants in at 73 centers. An additional 34 centers had no screening activities, but received study medication; and an additional 17 centers had at least 1 participant screened, but did not randomize any participants.
Pre-assignment Details: Participants enrolled who had documented rheumatoid arthritis with a duration of at least 3 months as determined by the investigator using standardly accepted criteria, had received methotrexate for at least 3 months to treat their rheumatoid arthritis, and were free of any signs or symptoms of infection.
Groups:
- PF-04171327 1 mg: Participants received PF-04171327 1 mg Once daily (QD) for 8 weeks. From week 9 through 10, the participants received 1 mg PF-04171327 + 1 placebo tablet every other day. From week 11 through 12, the participants received 1 mg PF-04171327 + 1 placebo tablet every 3 days.
- PF-04171327 5 mg: Participants received PF-04171327 5 mg QD for 8 weeks. After 8 weeks of study treatment, participants were tapered off study drug. From week 9 through 10, the participants received 1 mg PF-04171327 + 1 placebo tablet every other day. From week 11 through 12, the participants received 1 mg PF-04171327 + 1 placebo tablet every 3 days.
- PF-04171327 10 mg: Participants received PF-04171327 10 mg QD for 8 weeks. After 8 weeks of study treatment, participants were tapered off study drug. From week 9 through 10, the participants received 1 mg PF-04171327 + 1 placebo tablet every other day. From week 11 through 12, the participants received 1 mg PF-04171327 + 1 placebo tablet every 3 days.
- PF-04171327 15 mg: Participants received PF-04171327 15 mg QD for 8 weeks. After 8 weeks of study treatment, participants were tapered off study drug. From week 9 through 10, the participants received 1 mg PF-04171327 + 1 placebo tablet every other day. From week 11 through 12, the participants received 1 mg PF-04171327 + 1 placebo tablet every 3 days.
- Prednisone 5 mg: Participants received prednisone 5 mg QD for 8 weeks. From week 9 through 10, the participants received 1 prednisone 5 mg tablet + 1 placebo tablet every other day. From week 11 through 12, the participants received 1 prednisone 5 mg tablet + 1 placebo tablet every 3 days.
- Prednisone 10 mg: Participants received prednisone 10 mg QD for 8 weeks. After 8 weeks of treatment, participants were tapered off prednisone dosage. From week 9 through 10, the participants received 1 prednisone 5 mg tablet + 1 placebo tablet every other day. From week 11 through 12, the participants received 1 prednisone 5 mg tablet + 1 placebo tablet every 3 days.
- Placebo: Participants received placebo QD until week 12.
Period: Overall Study
Arm/Group | PF-04171327 1 mg | PF-04171327 5 mg | PF-04171327 10 mg | PF-04171327 15 mg | Prednisone 5 mg | Prednisone 10 mg | Placebo
Started | 45 | 47 | 45 | 48 | 45 | 46 | 47
Completed | 42 | 40 | 44 | 43 | 44 | 44 | 39
Not Completed | 3 | 7 | 1 | 5 | 1 | 2 | 8
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Other | 0 | 2 | 0 | 2 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Medication error without associated AE | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 2 | 3 | 1 | 2 | 0 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-04171327 1 mg | PF-04171327 5 mg | PF-04171327 10 mg | PF-04171327 15 mg | Prednisone 5 mg | Prednisone 10 mg | Placebo | Total
Number analyzed (Participants) | 45 | 47 | 45 | 48 | 45 | 46 | 47 | 323
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.4 (14.2) | 55.1 (12.1) | 54.7 (13.1) | 54.0 (11.1) | 52.9 (11.2) | 57.3 (10.7) | 55.2 (13.2) | 54.3 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 38 | 34 | 37 | 39 | 41 | 37 | 259
  Male | 12 | 9 | 11 | 11 | 6 | 5 | 10 | 64

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a 20% Improvement in American College of Rheumatology (ACR) Criteria at Week 8
Description: ACR20 response: greater than or equal to (≥) 20 percent (%) improvement in tender joint count; ≥ 20% improvement in swollen joint count; and ≥ 20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP).
Time Frame: Week 8
Population: Full Analysis Set (FAS) included all participants who were randomized to the study and received at least one dose of the randomized study drug (PF 04171327, prednisone, or placebo). N= number of participants with observations.
Measure: Number; unit: Percentage of participants
Arm/Group | PF-04171327 1 mg | PF-04171327 5 mg | PF-04171327 10 mg | PF-04171327 15 mg | Prednisone 5 mg | Prednisone 10 mg | Placebo
Number analyzed (Participants) | 45 | 47 | 45 | 48 | 45 | 46 | 47
Percentage of participants | 47 | 61 | 69 | 73 | 51 | 71 | 37
Statistical Analysis 1: Comparison: PF-04171327 1 mg vs Placebo; Bayesian 4 Parameter Emax Model Based Estimates are provided; Test type: Superiority or Other; Mean Difference (Final Values) = 10, 60% CI 2-sided [5 to 15] — Superiority criterion versus placebo: Lower bound of 60% credible interval >20%. Non-responder imputation was used to handle dropouts at Week 8
Statistical Analysis 2: Comparison: PF-04171327 5 mg vs Placebo; Bayesian 4 Parameter Emax Model Based Estimates are provided; Test type: Superiority or Other; Mean Difference (Final Values) = 24, 60% CI 2-sided [18 to 31] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: PF-04171327 10 mg vs Placebo; Bayesian 4 Parameter Emax Model Based Estimates are provided; Test type: Superiority or Other; Mean Difference (Final Values) = 32, 60% CI 2-sided [25 to 39] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: PF-04171327 15 mg vs Placebo; Bayesian 4 Parameter Emax Model Based Estimates are provided; Test type: Superiority or Other; Mean Difference (Final Values) = 36, 60% CI 2-sided [29 to 43] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Prednisone 5 mg vs Placebo; Bayesian 4 Parameter Emax Model Based Estimates are provided; Test type: Superiority or Other; Mean Difference (Final Values) = 14, 60% CI 2-sided [6 to 22] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Prednisone 10 mg vs Placebo; Bayesian 4 Parameter Emax Model Based Estimates are provided; Test type: Superiority or Other; Mean Difference (Final Values) = 34, 60% CI 2-sided [27 to 42] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; Bayesian 4 Parameter Emax Model Based Estimates are provided; Test type: Superiority or Other; Mean Difference (Final Values) = -24, 60% CI 2-sided [-32 to -17] — Non inferiority criterion versus prednisone 10 mg: Lower bound of 60% credible interval >-5%. Non-responder imputation was used to handle dropouts at Week 8
Statistical Analysis 8: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; Bayesian 4 Parameter Emax Model Based Estimates are provided; Test type: Superiority or Other; Mean Difference (Final Values) = -10, 60% CI 2-sided [-16 to -4] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 9: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; Bayesian 4 Parameter Emax Model Based Estimates are provided; Test type: Superiority or Other; Mean Difference (Final Values) = -2, 60% CI 2-sided [-9 to 4] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 10: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; Bayesian 4 Parameter Emax Model Based Estimates are provided; Test type: Superiority or Other; Mean Difference (Final Values) = 1, 60% CI 2-sided [-5 to 8] — [estimate comment as in outcome 1, analysis 7]

2. Primary Outcome: Mean Percent Change From Baseline in 0 Hour Procollagen Type 1 N Terminal Propeptide (P1NP) at Week 8 (Comparisons to Prednisone 5 mg)
Description: Change from baseline in P1NP at week 8 is presented in this outcome measure.
Time Frame: Week 8
Population: FAS included all participants who were randomized to the study and received at least one dose of the randomized study drug (PF 04171327, prednisone, or placebo). N= number of participants with observations.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | PF-04171327 1 mg | PF-04171327 5 mg | PF-04171327 10 mg | PF-04171327 15 mg | Prednisone 5 mg | Prednisone 10 mg | Placebo
Number analyzed (Participants) | 44 | 42 | 44 | 43 | 43 | 44 | 41
Percent change | -3.25 (5.50) | -11.60 (5.55) | -9.96 (5.49) | -16.63 (5.55) | -4.89 (5.55) | -20.14 (5.50) | 14.19 (5.56)
Statistical Analysis 1: Comparison: PF-04171327 1 mg vs Prednisone 5 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 1.64, 95% CI 2-sided [-13.75 to 17.03] — Statistical analysis was performed using a repeated measures mixed model with fixed effects for treatment and visit, treatment by visit interaction and baseline value; unstructured covariance matrix was used
Statistical Analysis 2: Comparison: PF-04171327 5 mg vs Prednisone 5 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -6.71, 90% CI 2-sided [-22.16 to 8.75] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: PF-04171327 10 mg vs Prednisone 5 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -5.07, 90% CI 2-sided [-20.45 to 10.30] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: PF-04171327 15 mg vs Prednisone 5 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -11.74, 90% CI 2-sided [-27.19 to 3.72] — [estimate comment as in outcome 2, analysis 1]

3. Primary Outcome: Mean Percent Change From Baseline in 0 Hour Urinary N Telopeptide/Urinary Creatinine (uNTx/uCr) at Week 8 (Comparisons to Prednisone 5 mg)
Description: Change from baseline in uNTx/uCr at week 8 is presented in this outcome measure.
Time Frame: Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | PF-04171327 1 mg | PF-04171327 5 mg | PF-04171327 10 mg | PF-04171327 15 mg | Prednisone 5 mg | Prednisone 10 mg | Placebo
Number analyzed (Participants) | 43 | 42 | 43 | 43 | 43 | 43 | 42
Percent change | 6.08 (5.83) | -3.78 (5.88) | 6.96 (5.86) | 15.57 (5.83) | 2.74 (5.87) | -9.14 (5.83) | 3.81 (5.88)
Statistical Analysis 1: Comparison: PF-04171327 1 mg vs Prednisone 5 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 3.34, 95% CI 2-sided [-12.92 to 19.61] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: PF-04171327 5 mg vs Prednisone 5 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -6.52, 90% CI 2-sided [-22.86 to 9.81] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: PF-04171327 10 mg vs Prednisone 5 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 4.22, 90% CI 2-sided [-12.11 to 20.55] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: PF-04171327 15 mg vs Prednisone 5 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 12.83, 90% CI 2-sided [-3.49 to 29.15] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Percentage of Participants Achieving ACR20 Response at Weeks 2, 4, and 12 (Comparisons to Placebo, and Prednisone 10 mg)
Description: ACR20 response: greater than or equal to (≥) 90 percent (%) improvement in tender or swollen joint counts and 90% improvement in 3 of the following 5 criteria: 1) physician's global assessment of disease activity, 2) participant's assessment of disease activity, 3) participant's assessment of pain, 4) participant's assessment of functional disability via a health assessment questionnaire, and 5) C-reactive protein at each visit.
Time Frame: Weeks 2, 4, and 12 (taper period)
Population: FAS included all participants who were randomized to the study and received at least one dose of the randomized study drug (PF 04171327, prednisone, or placebo). Note, N = number of participants in FAS and n = number of participants with observations in the below table.
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-04171327 1 mg | PF-04171327 5 mg | PF-04171327 10 mg | PF-04171327 15 mg | Prednisone 5 mg | Prednisone 10 mg | Placebo
Number analyzed (Participants) | 45 | 47 | 45 | 48 | 45 | 46 | 47
Percentage of Participants
  Week 2: number analyzed (Participants) | 44 | 46 | 45 | 47 | 45 | 46 | 44
  Week 2 | 31.82 (7.02) | 32.61 (6.91) | 40.00 (7.30) | 42.55 (7.21) | 28.89 (6.75) | 36.96 (7.11) | 20.45 (6.08)
  Week 4: number analyzed (Participants) | 45 | 47 | 45 | 47 | 45 | 46 | 45
  Week 4 | 31.11 (6.90) | 55.32 (7.25) | 66.67 (7.02) | 53.19 (7.27) | 48.89 (7.45) | 65.22 (7.02) | 40.00 (7.30)
  Week 12: number analyzed (Participants) | 45 | 47 | 45 | 47 | 45 | 46 | 45
  Week 12 | 35.56 (7.13) | 48.94 (7.29) | 55.56 (7.40) | 38.30 (7.09) | 48.89 (7.45) | 56.52 (7.30) | 33.33 (7.02)
Statistical Analysis 1: Comparison: PF-04171327 1 mg vs Placebo; Week 2 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 11.36, 95% CI 2-sided [-6.84 to 29.56] — Non-responder imputation was used to handle dropouts
Statistical Analysis 2: Comparison: PF-04171327 5 mg vs Placebo; Week 2 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 12.15, 95% CI 2-sided [-5.88 to 30.19] — Non-responder imputation was used to handle dropouts
Statistical Analysis 3: Comparison: PF-04171327 10 mg vs Placebo; Week 2 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 19.54, 95% CI 2-sided [0.91 to 38.17] — Non-responder imputation was used to handle dropouts
Statistical Analysis 4: Comparison: PF-04171327 15 mg vs Placebo; Week 2 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 22.09, 95% CI 2-sided [3.60 to 40.58] — Non-responder imputation was used to handle dropouts
Statistical Analysis 5: Comparison: Prednisone 5 mg vs Placebo; Week 2 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 8.43, 95% CI 2-sided [-9.38 to 26.25] — Non-responder imputation was used to handle dropouts
Statistical Analysis 6: Comparison: Prednisone 10 mg vs Placebo; Week 2 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 16.50, 95% CI 2-sided [-1.84 to 34.84] — Non-responder imputation was used to handle dropouts
Statistical Analysis 7: Comparison: PF-04171327 1 mg vs Placebo; Week 4 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = -8.88, 95% CI 2-sided [-28.58 to 10.80] — Non-responder imputation was used to handle dropouts
Statistical Analysis 8: Comparison: PF-04171327 5 mg vs Placebo; Week 4 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 15.31, 95% CI 2-sided [-4.85 to 35.49] — Non-responder imputation was used to handle dropouts
Statistical Analysis 9: Comparison: PF-04171327 10 mg vs Placebo; Week 4 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 26.66, 95% CI 2-sided [6.80 to 46.53] — Non-responder imputation was used to handle dropouts
Statistical Analysis 10: Comparison: PF-04171327 15 mg vs Placebo; Week 4 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 13.19, 95% CI 2-sided [-7.01 to 33.40] — Non-responder imputation was used to handle dropouts
Statistical Analysis 11: Comparison: Prednisone 5 mg vs Placebo; Week 4 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 8.88, 95% CI 2-sided [-11.56 to 29.33] — Non-responder imputation was used to handle dropouts
Statistical Analysis 12: Comparison: Prednisone 10 mg vs Placebo; Week 4 comparisons presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 25.21, 95% CI 2-sided [5.35 to 45.07] — Non-responder imputation was used to handle dropouts
Statistical Analysis 13: Comparison: PF-04171327 1 mg vs Placebo; Week 12 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 2.22, 95% CI 2-sided [-17.40 to 21.85] — Non-responder imputation was used to handle dropouts
Statistical Analysis 14: Comparison: PF-04171327 5 mg vs Placebo; Week 12 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 15.60, 95% CI 2-sided [-4.24 to 35.45] — Non-responder imputation was used to handle dropouts
Statistical Analysis 15: Comparison: PF-04171327 10 mg vs Placebo; Week 12 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 22.22, 95% CI 2-sided [2.20 to 42.23] — Non-responder imputation was used to handle dropouts
Statistical Analysis 16: Comparison: PF-04171327 15 mg vs Placebo; Week 12 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 4.96, 95% CI 2-sided [-14.60 to 24.53] — Non-responder imputation was used to handle dropouts
Statistical Analysis 17: Comparison: Prednisone 5 mg vs Placebo; Week 12 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 15.55, 95% CI 2-sided [-4.51 to 35.63] — Non-responder imputation was used to handle dropouts
Statistical Analysis 18: Comparison: Prednisone 10 mg vs Placebo; Week 12 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 23.18, 95% CI 2-sided [3.31 to 43.06] — Non-responder imputation was used to handle dropouts
Statistical Analysis 19: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; Week 2 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = -5.13, 95% CI 2-sided [-24.73 to 14.45] — Non-responder imputation was used to handle dropouts
Statistical Analysis 20: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; Week 2 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = -4.34, 95% CI 2-sided [-23.79 to 15.09] — Non-responder imputation was used to handle dropouts
Statistical Analysis 21: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; Week 2 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = 3.04, 95% CI 2-sided [-16.94 to 23.02] — Non-responder imputation was used to handle dropouts
Statistical Analysis 22: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; Week 2 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = 5.59, 95% CI 2-sided [-14.26 to 25.45] — Non-responder imputation was used to handle dropouts
Statistical Analysis 23: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; Week 4 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = -34.10, 95% CI 2-sided [-53.40 to -14.80] — Non-responder imputation was used to handle dropouts
Statistical Analysis 24: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; Week 4 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = -9.89, 95% CI 2-sided [-29.68 to 9.88] — Non-responder imputation was used to handle dropouts
Statistical Analysis 25: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; Week 4 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = 1.44, 95% CI 2-sided [-18.02 to 20.92] — Non-responder imputation was used to handle dropouts
Statistical Analysis 26: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; Week 4 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = -12.02, 95% CI 2-sided [-31.84 to 7.79] — Non-responder imputation was used to handle dropouts
Statistical Analysis 27: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; Week 12 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = -20.96, 95% CI 2-sided [-40.98 to -0.94] — Non-responder imputation was used to handle dropouts
Statistical Analysis 28: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; Week 12 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = -7.58, 95% CI 2-sided [-27.82 to 12.65] — Non-responder imputation was used to handle dropouts
Statistical Analysis 29: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; Week 12 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = -0.96, 95% CI 2-sided [-21.36 to 19.43] — Non-responder imputation was used to handle dropouts
Statistical Analysis 30: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; Week 12 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = -18.22, 95% CI 2-sided [-38.18 to 1.73] — Non-responder imputation was used to handle dropouts

5. Secondary Outcome: Percentage of Participants Achieving ACR50 Response at Weeks 2, 4, 6, 8 and 12 (Comparisons to Placebo, and Prednisone 10 mg)
Description: ACR50 response: greater than or equal to (≥) 50 percent (%) improvement in tender or swollen joint counts and 50% improvement in 3 of the following 5 criteria: 1) physician's global assessment of disease activity, 2) participant's assessment of disease activity, 3) participant's assessment of pain, 4) participant's assessment of functional disability via a health assessment questionnaire, and 5) C-reactive protein at each visit.
Time Frame: Weeks 2, 4, 6, 8, and 12 (taper period)
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-04171327 1 mg | PF-04171327 5 mg | PF-04171327 10 mg | PF-04171327 15 mg | Prednisone 5 mg | Prednisone 10 mg | Placebo
Number analyzed (Participants) | 45 | 47 | 45 | 48 | 45 | 46 | 47
Percentage of Participants
  Week 2: number analyzed (Participants) | 44 | 46 | 45 | 47 | 45 | 46 | 44
  Week 2 | 4.55 (3.14) | 8.70 (4.15) | 8.89 (4.24) | 25.53 (6.36) | 2.22 (2.19) | 19.57 (5.84) | 6.82 (3.79)
  Week 4: number analyzed (Participants) | 45 | 47 | 45 | 47 | 45 | 46 | 45
  Week 4 | 8.89 (4.24) | 23.40 (6.17) | 35.56 (7.13) | 27.66 (6.52) | 11.11 (4.68) | 30.43 (6.78) | 11.11 (4.68)
  Week 6: number analyzed (Participants) | 45 | 47 | 45 | 47 | 45 | 46 | 45
  Week 6 | 11.11 (4.68) | 27.66 (6.52) | 40.00 (7.30) | 42.55 (7.21) | 24.44 (6.40) | 36.96 (7.11) | 15.56 (5.40)
  Week 8: number analyzed (Participants) | 45 | 47 | 45 | 47 | 45 | 46 | 45
  Week 8 | 22.22 (6.19) | 31.91 (6.79) | 48.89 (7.45) | 42.55 (7.21) | 26.67 (6.59) | 45.65 (7.34) | 13.33 (5.16)
  Week 12: number analyzed (Participants) | 45 | 47 | 45 | 47 | 45 | 46 | 45
  Week 12 | 17.78 (5.69) | 21.28 (5.96) | 24.44 (6.40) | 17.02 (5.48) | 26.67 (6.59) | 23.91 (6.28) | 17.78 (5.69)
Statistical Analysis 1: Comparison: PF-04171327 1 mg vs Placebo; Week 2 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = -2.27, 95% CI 2-sided [-11.93 to 7.38] — Non-responder imputation was used to handle dropouts
Statistical Analysis 2: Comparison: PF-04171327 5 mg vs Placebo; Week 2 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 1.87, 95% CI 2-sided [-9.15 to 12.91] — Non-responder imputation was used to handle dropouts
Statistical Analysis 3: Comparison: PF-04171327 10 mg vs Placebo; Week 2 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 2.07, 95% CI 2-sided [-9.09 to 13.23] — Non-responder imputation was used to handle dropouts
Statistical Analysis 4: Comparison: PF-04171327 15 mg vs Placebo; Week 2 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 18.71, 95% CI 2-sided [4.19 to 33.23] — Non-responder imputation was used to handle dropouts
Statistical Analysis 5: Comparison: Prednisone 5 mg vs Placebo; Week 2 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = -4.59, 95% CI 2-sided [-13.19 to 4.00] — Non-responder imputation was used to handle dropouts
Statistical Analysis 6: Comparison: Prednisone 10 mg vs Placebo; Week 2 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 12.74, 95% CI 2-sided [-0.92 to 26.41] — Non-responder imputation was used to handle dropouts
Statistical Analysis 7: Comparison: PF-04171327 1 mg vs Placebo; Week 4 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = -2.22, 95% CI 2-sided [-14.60 to 10.16] — Non-responder imputation was used to handle dropouts
Statistical Analysis 8: Comparison: PF-04171327 5 mg vs Placebo; Week 4 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 12.29, 95% CI 2-sided [-2.90 to 27.48] — Non-responder imputation was used to handle dropouts
Statistical Analysis 9: Comparison: PF-04171327 10 mg vs Placebo; Week 4 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 24.44, 95% CI 2-sided [7.71 to 41.17] — Non-responder imputation was used to handle dropouts
Statistical Analysis 10: Comparison: PF-04171327 15 mg vs Placebo; Week 4 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 16.54, 95% CI 2-sided [0.80 to 32.29] — Non-responder imputation was used to handle dropouts
Statistical Analysis 11: Comparison: Prednisone 5 mg vs Placebo; Week 4 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 0.0, 95% CI 2-sided [-12.98 to 12.98] — Non-responder imputation was used to handle dropouts
Statistical Analysis 12: Comparison: Prednisone 10 mg vs Placebo; Week 4 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 19.32, 95% CI 2-sided [3.16 to 35.48] — Non-responder imputation was used to handle dropouts
Statistical Analysis 13: Comparison: PF-04171327 1 mg vs Placebo; Week 6 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = -4.44, 95% CI 2-sided [-18.46 to 9.57] — Non-responder imputation was used to handle dropouts
Statistical Analysis 14: Comparison: PF-04171327 5 mg vs Placebo; Week 6 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 12.10, 95% CI 2-sided [-4.49 to 28.70] — Non-responder imputation was used to handle dropouts
Statistical Analysis 15: Comparison: PF-04171327 10 mg vs Placebo; Week 6 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 24.44, 95% CI 2-sided [6.63 to 42.24] — Non-responder imputation was used to handle dropouts
Statistical Analysis 16: Comparison: PF-04171327 15 mg vs Placebo; Week 6 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 26.99, 95% CI 2-sided [9.33 to 44.65] — Non-responder imputation was used to handle dropouts
Statistical Analysis 17: Comparison: Prednisone 5 mg vs Placebo; Week 6 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 8.88, 95% CI 2-sided [-7.53 to 25.31] — Non-responder imputation was used to handle dropouts
Statistical Analysis 18: Comparison: Prednisone 10 mg vs Placebo; Week 6 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 21.40, 95% CI 2-sided [3.88 to 38.91] — Non-responder imputation was used to handle dropouts
Statistical Analysis 19: Comparison: PF-04171327 1 mg vs Placebo; Week 8 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 8.88, 95% CI 2-sided [-6.80 to 24.57] — Non-responder imputation was used to handle dropouts
Statistical Analysis 20: Comparison: PF-04171327 5 mg vs Placebo; Week 8 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 18.58, 95% CI 2-sided [1.96 to 35.20] — Non-responder imputation was used to handle dropouts
Statistical Analysis 21: Comparison: PF-04171327 10 mg vs Placebo; Week 8 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 35.55, 95% CI 2-sided [17.89 to 53.21] — Non-responder imputation was used to handle dropouts
Statistical Analysis 22: Comparison: PF-04171327 15 mg vs Placebo; Week 8 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 29.21, 95% CI 2-sided [11.94 to 46.49] — Non-responder imputation was used to handle dropouts
Statistical Analysis 23: Comparison: Prednisone 5 mg vs Placebo; Week 8 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 13.33, 95% CI 2-sided [-2.96 to 29.63] — Non-responder imputation was used to handle dropouts
Statistical Analysis 24: Comparison: Prednisone 10 mg vs Placebo; Week 8 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 32.31, 95% CI 2-sided [14.83 to 49.80] — Non-responder imputation was used to handle dropouts
Statistical Analysis 25: Comparison: PF-04171327 1 mg vs Placebo; Week 12 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 0.00, 95% CI 2-sided [-15.79 to 15.79] — Non-responder imputation was used to handle dropouts
Statistical Analysis 26: Comparison: PF-04171327 5 mg vs Placebo; Week 12 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 3.49, 95% CI 2-sided [-12.67 to 19.67] — Non-responder imputation was used to handle dropouts
Statistical Analysis 27: Comparison: PF-04171327 10 mg vs Placebo; Week 12 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 6.66, 95% CI 2-sided [-10.13 to 23.47] — Non-responder imputation was used to handle dropouts
Statistical Analysis 28: Comparison: PF-04171327 15 mg vs Placebo; Week 12 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = -0.75, 95% CI 2-sided [-16.25 to 14.74] — Non-responder imputation was used to handle dropouts
Statistical Analysis 29: Comparison: Prednisone 5 mg vs Placebo; Week 12 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 8.88, 95% CI 2-sided [-8.19 to 25.96] — Non-responder imputation was used to handle dropouts
Statistical Analysis 30: Comparison: Prednisone 10 mg vs Placebo; Week 12 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 6.13, 95% CI 2-sided [-10.50 to 22.77] — Non-responder imputation was used to handle dropouts
Statistical Analysis 31: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; Week 2 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = -15.01, 95% CI 2-sided [-28.03 to -2.00] — Non-responder imputation was used to handle dropouts
Statistical Analysis 32: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; Week 2 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = -10.86, 95% CI 2-sided [-24.93 to 3.19] — Non-responder imputation was used to handle dropouts
Statistical Analysis 33: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; Week 2 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = -10.67, 95% CI 2-sided [-24.83 to 3.48] — Non-responder imputation was used to handle dropouts
Statistical Analysis 34: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; Week 2 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = 5.96, 95% CI 2-sided [-10.96 to 22.90] — Non-responder imputation was used to handle dropouts
Statistical Analysis 35: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; Week 4 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = -21.54, 95% CI 2-sided [-37.22 to -5.86] — Non-responder imputation was used to handle dropouts
Statistical Analysis 36: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; Week 4 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = -7.03, 95% CI 2-sided [-25.01 to 10.95] — Non-responder imputation was used to handle dropouts
Statistical Analysis 37: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; Week 4 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = 5.12, 95% CI 2-sided [-14.17 to 24.41] — Non-responder imputation was used to handle dropouts
Statistical Analysis 38: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; Week 4 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = -2.77, 95% CI 2-sided [-21.22 to 15.67] — Non-responder imputation was used to handle dropouts
Statistical Analysis 39: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; Week 6 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = -25.84, 95% CI 2-sided [-42.54 to -9.14] — Non-responder imputation was used to handle dropouts
Statistical Analysis 40: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; Week 6 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = -9.29, 95% CI 2-sided [-28.22 to 9.62] — Non-responder imputation was used to handle dropouts
Statistical Analysis 41: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; Week 6 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = 3.04, 95% CI 2-sided [-16.94 to 23.02] — Non-responder imputation was used to handle dropouts
Statistical Analysis 42: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; Week 6 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = 5.59, 95% CI 2-sided [-14.26 to 25.45] — Non-responder imputation was used to handle dropouts
Statistical Analysis 43: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; Week 8 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = -23.42, 95% CI 2-sided [-42.26 to -4.59] — Non-responder imputation was used to handle dropouts
Statistical Analysis 44: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; Week 8 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = -13.73, 95% CI 2-sided [-33.35 to 5.87] — Non-responder imputation was used to handle dropouts
Statistical Analysis 45: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; Week 8 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = 3.23, 95% CI 2-sided [-17.26 to 23.74] — Non-responder imputation was used to handle dropouts
Statistical Analysis 46: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; Week 8 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = -3.09, 95% CI 2-sided [-23.27 to 17.07] — Non-responder imputation was used to handle dropouts
Statistical Analysis 47: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; Week 12 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = -6.13, 95% CI 2-sided [-22.77 to 10.50] — Non-responder imputation was used to handle dropouts
Statistical Analysis 48: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; Week 12 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = -2.63, 95% CI 2-sided [-19.63 to 14.35] — Non-responder imputation was used to handle dropouts
Statistical Analysis 49: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; Week 12 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = 0.53, 95% CI 2-sided [-17.06 to 18.12] — Non-responder imputation was used to handle dropouts
Statistical Analysis 50: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; Week 12 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = -6.89, 95% CI 2-sided [-23.24 to 9.46] — Non-responder imputation was used to handle dropouts

6. Secondary Outcome: Percentage of Participants Achieving ACR70 Response at Weeks 2, 4, 6, 8 and 12 (Comparisons to Placebo, and Prednisone 10 mg)
Description: ACR70 response: greater than or equal to (≥) 70 percent (%) improvement in tender or swollen joint counts and 70% improvement in 3 of the following 5 criteria: 1) physician's global assessment of disease activity, 2) subject's assessment of disease activity, 3) subject's assessment of pain, 4) subject's assessment of functional disability via a health assessment questionnaire, and 5) C-reactive protein at each visit.
Time Frame: Weeks 2, 4, 6, 8, and 12 (taper period)
Population: Full analysis set was used. Note, N = number of participants in FAS and n = number of participants with observations in the below table.
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-04171327 1 mg | PF-04171327 5 mg | PF-04171327 10 mg | PF-04171327 15 mg | Prednisone 5 mg | Prednisone 10 mg | Placebo
Number analyzed (Participants) | 45 | 47 | 45 | 48 | 45 | 46 | 47
Percentage of Participants
  Week 2: number analyzed (Participants) | 44 | 46 | 45 | 47 | 45 | 46 | 44
  Week 2 | 0.0 | 4.35 | 2.22 | 6.38 | 2.22 | 8.70 | 0.0
  Week 4: number analyzed (Participants) | 45 | 47 | 45 | 47 | 45 | 46 | 45
  Week 4 | 0.0 | 8.51 | 15.56 | 17.02 | 4.44 | 15.22 | 0.0
  Week 6: number analyzed (Participants) | 45 | 47 | 45 | 47 | 45 | 46 | 45
  Week 6 | 2.22 | 12.77 | 13.33 | 17.02 | 6.67 | 21.74 | 4.44
  Week 8: number analyzed (Participants) | 45 | 47 | 45 | 47 | 45 | 46 | 45
  Week 8 | 8.89 | 17.02 | 26.67 | 21.28 | 6.67 | 26.09 | 11.11
  Week 12: number analyzed (Participants) | 45 | 47 | 45 | 47 | 45 | 46 | 45
  Week 12 | 6.67 | 12.77 | 6.67 | 8.51 | 11.11 | 10.87 | 6.67
Statistical Analysis 1: Comparison: PF-04171327 1 mg vs Placebo; Week 2 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 0.00, 95% CI 2-sided [0.00 to 0.00] — Non-responder imputation was used to handle dropouts
Statistical Analysis 2: Comparison: PF-04171327 5 mg vs Placebo; Week 2 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 4.34, 95% CI 2-sided [-1.54 to 10.24] — Non-responder imputation was used to handle dropouts
Statistical Analysis 3: Comparison: PF-04171327 10 mg vs Placebo; Week 2 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 2.22, 95% CI 2-sided [-2.08 to 6.52] — Non-responder imputation was used to handle dropouts
Statistical Analysis 4: Comparison: PF-04171327 15 mg vs Placebo; Week 2 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 6.38, 95% CI 2-sided [-0.60 to 13.37] — Non-responder imputation was used to handle dropouts
Statistical Analysis 5: Comparison: Prednisone 5 mg vs Placebo; Week 2 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 2.22, 95% CI 2-sided [-2.08 to 6.52] — Non-responder imputation was used to handle dropouts
Statistical Analysis 6: Comparison: Prednisone 10 mg vs Placebo; Week 2 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 8.69, 95% CI 2-sided [0.55 to 16.83] — Non-responder imputation was used to handle dropouts
Statistical Analysis 7: Comparison: PF-04171327 1 mg vs Placebo; Week 4 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 0.00, 95% CI 2-sided [0.00 to 0.00] — Non-responder imputation was used to handle dropouts
Statistical Analysis 8: Comparison: PF-04171327 5 mg vs Placebo; Week 4 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 8.51, 95% CI 2-sided [0.53 to 16.48] — Non-responder imputation was used to handle dropouts
Statistical Analysis 9: Comparison: PF-04171327 10 mg vs Placebo; Week 4 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 15.55, 95% CI 2-sided [4.96 to 26.14] — Non-responder imputation was used to handle dropouts
Statistical Analysis 10: Comparison: PF-04171327 15 mg vs Placebo; Week 4 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 17.02, 95% CI 2-sided [6.27 to 27.76] — Non-responder imputation was used to handle dropouts
Statistical Analysis 11: Comparison: Prednisone 5 mg vs Placebo; Week 4 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 4.44, 95% CI 2-sided [-1.57 to 10.46] — Non-responder imputation was used to handle dropouts
Statistical Analysis 12: Comparison: Prednisone 10 mg vs Placebo; Week 4 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 15.21, 95% CI 2-sided [4.83 to 25.59] — Non-responder imputation was used to handle dropouts
Statistical Analysis 13: Comparison: PF-04171327 1 mg vs Placebo; Week 6 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = -2.22, 95% CI 2-sided [-9.62 to 5.18] — Non-responder imputation was used to handle dropouts
Statistical Analysis 14: Comparison: PF-04171327 5 mg vs Placebo; Week 6 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 8.32, 95% CI 2-sided [-2.96 to 19.60] — Non-responder imputation was used to handle dropouts
Statistical Analysis 15: Comparison: PF-04171327 10 mg vs Placebo; Week 6 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 8.88, 95% CI 2-sided [-2.72 to 20.50] — Non-responder imputation was used to handle dropouts
Statistical Analysis 16: Comparison: PF-04171327 15 mg vs Placebo; Week 6 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 12.57, 95% CI 2-sided [0.26 to 24.89] — Non-responder imputation was used to handle dropouts
Statistical Analysis 17: Comparison: Prednisone 5 mg vs Placebo; Week 6 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 2.22, 95% CI 2-sided [-7.23 to 11.67] — Non-responder imputation was used to handle dropouts
Statistical Analysis 18: Comparison: Prednisone 10 mg vs Placebo; Week 6 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 17.29, 95% CI 2-sided [3.94 to 30.64] — Non-responder imputation was used to handle dropouts
Statistical Analysis 19: Comparison: PF-04171327 1 mg vs Placebo; Week 8 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = -2.22, 95% CI 2-sided [-14.60 to 10.16] — Non-responder imputation was used to handle dropouts
Statistical Analysis 20: Comparison: PF-04171327 5 mg vs Placebo; Week 8 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 5.91, 95% CI 2-sided [-8.22 to 20.04] — Non-responder imputation was used to handle dropouts
Statistical Analysis 21: Comparison: PF-04171327 10 mg vs Placebo; Week 8 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 15.55, 95% CI 2-sided [-0.29 to 31.40] — Non-responder imputation was used to handle dropouts
Statistical Analysis 22: Comparison: PF-04171327 15 mg vs Placebo; Week 8 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 10.16, 95% CI 2-sided [-4.70 to 25.03] — Non-responder imputation was used to handle dropouts
Statistical Analysis 23: Comparison: Prednisone 5 mg vs Placebo; Week 8 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = -4.44, 95% CI 2-sided [-16.16 to 7.27] — Non-responder imputation was used to handle dropouts
Statistical Analysis 24: Comparison: Prednisone 10 mg vs Placebo; Week 8 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 14.97, 95% CI 2-sided [-0.68 to 30.63] — Non-responder imputation was used to handle dropouts
Statistical Analysis 25: Comparison: PF-04171327 1 mg vs Placebo; Week 12 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 0.00, 95% CI 2-sided [-10.30 to 10.30] — Non-responder imputation was used to handle dropouts
Statistical Analysis 26: Comparison: PF-04171327 5 mg vs Placebo; Week 12 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 6.09, 95% CI 2-sided [-5.90 to 18.10] — Non-responder imputation was used to handle dropouts
Statistical Analysis 27: Comparison: PF-04171327 10 mg vs Placebo; Week 12 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 0.00, 95% CI 2-sided [-10.30 to 10.30] — Non-responder imputation was used to handle dropouts
Statistical Analysis 28: Comparison: PF-04171327 15 mg vs Placebo; Week 12 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 1.84, 95% CI 2-sided [-8.96 to 12.64] — Non-responder imputation was used to handle dropouts
Statistical Analysis 29: Comparison: Prednisone 5 mg vs Placebo; Week 12 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 4.44, 95% CI 2-sided [-7.27 to 16.16] — Non-responder imputation was used to handle dropouts
Statistical Analysis 30: Comparison: Prednisone 10 mg vs Placebo; Week 12 analysis presented in this section for comparison to placebo; Test type: Superiority or Other; Difference in percentage = 4.20, 95% CI 2-sided [-7.37 to 15.77] — Non-responder imputation was used to handle dropouts
Statistical Analysis 31: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; Week 2 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = -8.69, 95% CI 2-sided [-16.83 to -0.55] — Non-responder imputation was used to handle dropouts
Statistical Analysis 32: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; Week 2 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = -4.34, 95% CI 2-sided [-14.39 to 5.70] — Non-responder imputation was used to handle dropouts
Statistical Analysis 33: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; Week 2 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = -6.47, 95% CI 2-sided [-15.68 to 2.73] — Non-responder imputation was used to handle dropouts
Statistical Analysis 34: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; Week 2 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = -2.31, 95% CI 2-sided [-13.04 to 8.41] — Non-responder imputation was used to handle dropouts
Statistical Analysis 35: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; Week 4 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = -15.21, 95% CI 2-sided [-25.59 to -4.83] — Non-responder imputation was used to handle dropouts
Statistical Analysis 36: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; Week 4 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = -6.70, 95% CI 2-sided [-19.79 to 6.38] — Non-responder imputation was used to handle dropouts
Statistical Analysis 37: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; Week 4 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = 0.33, 95% CI 2-sided [-14.49 to 15.16] — Non-responder imputation was used to handle dropouts
Statistical Analysis 38: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; Week 4 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = 1.80, 95% CI 2-sided [-13.13 to 16.74] — Non-responder imputation was used to handle dropouts
Statistical Analysis 39: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; Week 6 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = -19.51, 95% CI 2-sided [-32.19 to -6.84] — Non-responder imputation was used to handle dropouts
Statistical Analysis 40: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; Week 6 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = -8.97, 95% CI 2-sided [-24.24 to 6.29] — Non-responder imputation was used to handle dropouts
Statistical Analysis 41: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; Week 6 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = -8.40, 95% CI 2-sided [-23.92 to 7.10] — Non-responder imputation was used to handle dropouts
Statistical Analysis 42: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; Week 6 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = -4.71, 95% CI 2-sided [-20.76 to 11.32] — Non-responder imputation was used to handle dropouts
Statistical Analysis 43: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; Week 8 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = -17.19, 95% CI 2-sided [-32.36 to -2.02] — Non-responder imputation was used to handle dropouts
Statistical Analysis 44: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; Week 8 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = -9.06, 95% CI 2-sided [-25.69 to 7.56] — Non-responder imputation was used to handle dropouts
Statistical Analysis 45: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; Week 8 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = 0.57, 95% CI 2-sided [-17.53 to 18.68] — Non-responder imputation was used to handle dropouts
Statistical Analysis 46: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; Week 8 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = -4.81, 95% CI 2-sided [-22.07 to 12.45] — Non-responder imputation was used to handle dropouts
Statistical Analysis 47: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; Week 12 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = -4.20, 95% CI 2-sided [-15.77 to 7.37] — Non-responder imputation was used to handle dropouts
Statistical Analysis 48: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; Week 12 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = 1.89, 95% CI 2-sided [-11.21 to 15.00] — Non-responder imputation was used to handle dropouts
Statistical Analysis 49: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; Week 12 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = -4.20, 95% CI 2-sided [-15.77 to 7.37] — Non-responder imputation was used to handle dropouts
Statistical Analysis 50: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; Week 12 analysis presented in this section for comparison to prednisone 10 mg; Test type: Superiority or Other; Difference in percentage = -2.35, 95% CI 2-sided [-14.38 to 9.66] — Non-responder imputation was used to handle dropouts

7. Secondary Outcome: Change From Baseline in Tender-Joint Counts at Weeks 2, 4, 6, 8 (Comparisons to Placebo, and Prednisone 10 mg)
Description: Twenty-eight tender/painful joint count included the following joints: shoulders, elbows, wrists, metacarpophalangeal joints, proximal interphalangeal joints, and knees. Artificial joints were not assessed. These joints were assessed by a joint assessor, who was blinded to the participant's safety data, previous efficacy data and treatment randomization, to determine the number of joints that were considered tender or painful, and swollen.
Time Frame: Weeks 2, 4, 6, and 8
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Joints
Arm/Group | PF-04171327 1 mg | PF-04171327 5 mg | PF-04171327 10 mg | PF-04171327 15 mg | Prednisone 5 mg | Prednisone 10 mg | Placebo
Number analyzed (Participants) | 45 | 47 | 45 | 48 | 45 | 46 | 47
Joints
  Week 2: number analyzed (Participants) | 44 | 46 | 45 | 47 | 45 | 46 | 44
  Week 2 | -4.08 (0.74) | -5.55 (0.72) | -4.97 (0.73) | -5.65 (0.72) | -3.88 (0.73) | -5.38 (0.72) | -1.95 (0.74)
  Week 4: number analyzed (Participants) | 45 | 44 | 45 | 45 | 44 | 45 | 45
  Week 4 | -5.97 (0.80) | -6.99 (0.79) | -7.01 (0.80) | -6.93 (0.79) | -5.79 (0.80) | -7.44 (0.79) | -4.16 (0.80)
  Week 6: number analyzed (Participants) | 44 | 42 | 44 | 44 | 44 | 45 | 44
  Week 6 | -6.87 (0.87) | -8.83 (0.87) | -8.37 (0.87) | -8.31 (0.86) | -6.91 (0.87) | -8.75 (0.86) | -4.64 (0.87)
  Week 8: number analyzed (Participants) | 44 | 42 | 44 | 44 | 44 | 45 | 43
  Week 8 | -7.06 (0.91) | -8.65 (0.92) | -9.46 (0.91) | -9.17 (0.91) | -7.00 (0.91) | -8.84 (0.90) | -4.27 (0.92)
Statistical Analysis 1: Comparison: PF-04171327 1 mg vs Placebo; Week 2 analysis presented in this section for comparison to placebo. Statistical analyses presented are derived from mixed model with fixed effects for treatment, visit, treatment-by-visit interaction and baseline value; unstructured covariance matrix was used; Test type: Superiority or Other; Mean Difference (Final Values) = -2.13, 95% CI 2-sided [-4.19 to -0.07]
Statistical Analysis 2: Comparison: PF-04171327 5 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -3.60, 95% CI 2-sided [-5.63 to -1.57]
Statistical Analysis 3: Comparison: PF-04171327 10 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -3.02, 95% CI 2-sided [-5.06 to -0.97]
Statistical Analysis 4: Comparison: PF-04171327 15 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -3.70, 95% CI 2-sided [-5.73 to -1.68]
Statistical Analysis 5: Comparison: Prednisone 5 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -1.93, 95% CI 2-sided [-3.97 to 0.12]
Statistical Analysis 6: Comparison: Prednisone 10 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -3.43, 95% CI 2-sided [-5.46 to -1.39]
Statistical Analysis 7: Comparison: PF-04171327 1 mg vs Placebo; Week 4 analysis presented in this section for comparison to placebo. Statistical analyses presented are derived from mixed model with fixed effects for treatment, visit, treatment-by-visit interaction and baseline value; unstructured covariance matrix was used; Test type: Superiority or Other; Mean Difference (Final Values) = -1.81, 95% CI 2-sided [-4.03 to 0.42]
Statistical Analysis 8: Comparison: PF-04171327 5 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -2.83, 95% CI 2-sided [-5.04 to -0.62]
Statistical Analysis 9: Comparison: PF-04171327 10 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -2.85, 95% CI 2-sided [-5.07 to -0.64]
Statistical Analysis 10: Comparison: PF-04171327 15 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -2.77, 95% CI 2-sided [-4.98 to -0.56]
Statistical Analysis 11: Comparison: Prednisone 5 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -1.63, 95% CI 2-sided [-3.85 to 0.59]
Statistical Analysis 12: Comparison: Prednisone 10 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -3.27, 95% CI 2-sided [-5.48 to -1.06]
Statistical Analysis 13: Comparison: PF-04171327 1 mg vs Placebo; Week 6 analysis presented in this section for comparison to placebo. Statistical analyses presented are derived from mixed model with fixed effects for treatment, visit, treatment-by-visit interaction and baseline value; unstructured covariance matrix was used; Test type: Superiority or Other; Mean Difference (Final Values) = -2.23, 95% CI 2-sided [-4.66 to 0.20]
Statistical Analysis 14: Comparison: PF-04171327 5 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -4.19, 95% CI 2-sided [-6.62 to -1.77]
Statistical Analysis 15: Comparison: PF-04171327 10 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -3.73, 95% CI 2-sided [-6.15 to -1.31]
Statistical Analysis 16: Comparison: PF-04171327 15 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -3.68, 95% CI 2-sided [-6.09 to -1.26]
Statistical Analysis 17: Comparison: Prednisone 5 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -2.27, 95% CI 2-sided [-4.69 to 0.16]
Statistical Analysis 18: Comparison: Prednisone 10 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -4.11, 95% CI 2-sided [-6.52 to -1.70]
Statistical Analysis 19: Comparison: PF-04171327 1 mg vs Placebo; Week 8 analysis presented in this section for comparison to placebo. Statistical analyses presented are derived from mixed model with fixed effects for treatment, visit, treatment-by-visit interaction and baseline value; unstructured covariance matrix was used; Test type: Superiority or Other; Mean Difference (Final Values) = -2.80, 95% CI 2-sided [-5.34 to -0.25]
Statistical Analysis 20: Comparison: PF-04171327 5 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -4.38, 95% CI 2-sided [-6.93 to -1.83]
Statistical Analysis 21: Comparison: PF-04171327 10 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -5.20, 95% CI 2-sided [-7.74 to -2.66]
Statistical Analysis 22: Comparison: PF-04171327 15 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -4.90, 95% CI 2-sided [-7.43 to -2.36]
Statistical Analysis 23: Comparison: Prednisone 5 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -2.74, 95% CI 2-sided [-5.28 to -0.20]
Statistical Analysis 24: Comparison: Prednisone 10 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -4.57, 95% CI 2-sided [-7.10 to -2.05]
Statistical Analysis 25: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; Week 2 analysis presented in this section for comparison to prednisone 10 mg. Statistical analyses presented are derived from mixed model with fixed effects for treatment, visit, treatment-by-visit interaction and baseline value; unstructured covariance matrix was used; Test type: Superiority or Other; Mean Difference (Final Values) = 1.30, 95% CI 2-sided [-0.73 to 3.33]
Statistical Analysis 26: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 25]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-2.18 to 1.84]
Statistical Analysis 27: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 25]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.41, 95% CI 2-sided [-1.61 to 2.44]
Statistical Analysis 28: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 25]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.27, 95% CI 2-sided [-2.27 to 1.73]
Statistical Analysis 29: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; Week 4 analysis presented in this section for comparison to prednisone 10 mg. Statistical analyses presented are derived from mixed model with fixed effects for treatment, visit, treatment-by-visit interaction and baseline value; unstructured covariance matrix was used; Test type: Superiority or Other; Mean Difference (Final Values) = 1.47, 95% CI 2-sided [-0.74 to 3.68]
Statistical Analysis 30: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.45, 95% CI 2-sided [-1.76 to 2.65]
Statistical Analysis 31: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.42, 95% CI 2-sided [-1.79 to 2.63]
Statistical Analysis 32: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.51, 95% CI 2-sided [-1.69 to 2.70]
Statistical Analysis 33: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; Week 6 analysis presented in this section for comparison to prednisone 10 mg. Statistical analyses presented are derived from mixed model with fixed effects for treatment, visit, treatment-by-visit interaction and baseline value; unstructured covariance matrix was used; Test type: Superiority or Other; Mean Difference (Final Values) = 1.88, 95% CI 2-sided [-0.53 to 4.29]
Statistical Analysis 34: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 33]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-2.50 to 2.33]
Statistical Analysis 35: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 33]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.38, 95% CI 2-sided [-2.03 to 2.79]
Statistical Analysis 36: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 33]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.43, 95% CI 2-sided [-1.97 to 2.84]
Statistical Analysis 37: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; Week 8 analysis presented in this section for comparison to prednisone 10 mg. Statistical analyses presented are derived from mixed model with fixed effects for treatment, visit, treatment-by-visit interaction and baseline value; unstructured covariance matrix was used; Test type: Superiority or Other; Mean Difference (Final Values) = 1.78, 95% CI 2-sided [-0.75 to 4.30]
Statistical Analysis 38: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-2.34 to 2.73]
Statistical Analysis 39: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.62, 95% CI 2-sided [-3.14 to 1.89]
Statistical Analysis 40: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.33, 95% CI 2-sided [-2.84 to 2.19]

8. Secondary Outcome: Change From Baseline in Tender-Joint Counts at Week 12 (Descriptive Statistics)
Description: as for outcome 7
Time Frame: Week 12
Population: FAS included all participants who were randomized to the study and received at least one dose of the randomized study drug (PF 04171327, prednisone, or placebo). Note, N = number of participants with observations in the below table.
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | PF-04171327 1 mg | PF-04171327 5 mg | PF-04171327 10 mg | PF-04171327 15 mg | Prednisone 5 mg | Prednisone 10 mg | Placebo
Number analyzed (Participants) | 44 | 41 | 44 | 43 | 44 | 43 | 41
Joints | -6.25 (6.77) | -7.24 (6.13) | -6.16 (6.40) | -6.47 (7.54) | -7.07 (5.89) | -8.16 (4.66) | -5.59 (6.67)

9. Secondary Outcome: Change From Baseline in Swollen-Joint Counts at Weeks 2, 4, 6, and 8 (Comparisons to Placebo, and Prednisone 10 mg)
Description: as for outcome 7
Time Frame: Weeks 2, 4, 6, and 8
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Joints
Arm/Group | PF-04171327 1 mg | PF-04171327 5 mg | PF-04171327 10 mg | PF-04171327 15 mg | Prednisone 5 mg | Prednisone 10 mg | Placebo
Number analyzed (Participants) | 45 | 47 | 45 | 48 | 45 | 46 | 47
Joints
  Week 2: number analyzed (Participants) | 44 | 46 | 45 | 47 | 45 | 46 | 44
  Week 2 | -3.42 (0.62) | -4.70 (0.61) | -4.27 (0.62) | -5.36 (0.61) | -3.65 (0.62) | -5.04 (0.61) | -2.25 (0.62)
  Week 4: number analyzed (Participants) | 45 | 44 | 45 | 45 | 44 | 45 | 45
  Week 4 | -5.54 (0.70) | -5.85 (0.71) | -5.94 (0.70) | -7.00 (0.70) | -5.75 (0.71) | -6.71 (0.70) | -3.87 (0.70)
  Week 6: number analyzed (Participants) | 44 | 42 | 44 | 44 | 44 | 45 | 44
  Week 6 | -6.26 (0.69) | -6.90 (0.70) | -7.36 (0.69) | -7.68 (0.69) | -6.89 (0.69) | -8.02 (0.69) | -4.94 (0.69)
  Week 8: number analyzed (Participants) | 44 | 42 | 44 | 44 | 44 | 45 | 43
  Week 8 | -6.50 (0.79) | -7.45 (0.80) | -7.95 (0.79) | -7.83 (0.79) | -6.90 (0.79) | -8.38 (0.78) | -4.51 (0.80)
Statistical Analysis 1: Comparison: PF-04171327 1 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -1.18, 95% CI 2-sided [-2.91 to 0.56]
Statistical Analysis 2: Comparison: PF-04171327 5 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -2.45, 95% CI 2-sided [-4.17 to -0.73]
Statistical Analysis 3: Comparison: PF-04171327 10 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -2.03, 95% CI 2-sided [-3.76 to -0.29]
Statistical Analysis 4: Comparison: PF-04171327 15 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -3.11, 95% CI 2-sided [-4.82 to -1.40]
Statistical Analysis 5: Comparison: Prednisone 5 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -1.40, 95% CI 2-sided [-3.13 to 0.33]
Statistical Analysis 6: Comparison: Prednisone 10 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -2.80, 95% CI 2-sided [-4.52 to -1.07]
Statistical Analysis 7: Comparison: PF-04171327 1 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -1.67, 95% CI 2-sided [-3.63 to 0.29]
Statistical Analysis 8: Comparison: PF-04171327 5 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -1.98, 95% CI 2-sided [-3.94 to -0.01]
Statistical Analysis 9: Comparison: PF-04171327 10 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -2.07, 95% CI 2-sided [-4.03 to -0.11]
Statistical Analysis 10: Comparison: PF-04171327 15 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -3.13, 95% CI 2-sided [-5.09 to -1.17]
Statistical Analysis 11: Comparison: Prednisone 5 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -1.88, 95% CI 2-sided [-3.85 to 0.09]
Statistical Analysis 12: Comparison: Prednisone 10 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -2.84, 95% CI 2-sided [-4.79 to -0.88]
Statistical Analysis 13: Comparison: PF-04171327 1 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -1.32, 95% CI 2-sided [-3.25 to 0.60]
Statistical Analysis 14: Comparison: PF-04171327 5 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -1.97, 95% CI 2-sided [-3.90 to -0.04]
Statistical Analysis 15: Comparison: PF-04171327 10 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -2.43, 95% CI 2-sided [-4.35 to -0.50]
Statistical Analysis 16: Comparison: PF-04171327 15 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -2.75, 95% CI 2-sided [-4.66 to -0.83]
Statistical Analysis 17: Comparison: Prednisone 5 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -1.96, 95% CI 2-sided [-3.88 to -0.03]
Statistical Analysis 18: Comparison: Prednisone 10 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -3.08, 95% CI 2-sided [-5.00 to -1.17]
Statistical Analysis 19: Comparison: PF-04171327 1 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -1.99, 95% CI 2-sided [-4.20 to 0.21]
Statistical Analysis 20: Comparison: PF-04171327 5 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -2.95, 95% CI 2-sided [-5.17 to -0.72]
Statistical Analysis 21: Comparison: PF-04171327 10 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -3.44, 95% CI 2-sided [-5.65 to -1.23]
Statistical Analysis 22: Comparison: PF-04171327 15 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -3.32, 95% CI 2-sided [-5.52 to -1.12]
Statistical Analysis 23: Comparison: Prednisone 5 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -2.39, 95% CI 2-sided [-4.60 to -0.18]
Statistical Analysis 24: Comparison: Prednisone 10 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -3.87, 95% CI 2-sided [-6.07 to -1.68]
Statistical Analysis 25: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 25]; Test type: Superiority or Other; Mean Difference (Final Values) = 1.62, 95% CI 2-sided [-0.10 to 3.34]
Statistical Analysis 26: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 25]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.34, 95% CI 2-sided [-1.36 to 2.05]
Statistical Analysis 27: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 25]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.77, 95% CI 2-sided [-0.94 to 2.48]
Statistical Analysis 28: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 25]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.31, 95% CI 2-sided [-2.01 to 1.38]
Statistical Analysis 29: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = 1.17, 95% CI 2-sided [-0.79 to 3.12]
Statistical Analysis 30: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.86, 95% CI 2-sided [-1.10 to 2.82]
Statistical Analysis 31: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.76, 95% CI 2-sided [-1.19 to 2.72]
Statistical Analysis 32: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.29, 95% CI 2-sided [-2.24 to 1.66]
Statistical Analysis 33: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 33]; Test type: Superiority or Other; Mean Difference (Final Values) = 1.76, 95% CI 2-sided [-0.16 to 3.67]
Statistical Analysis 34: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 33]; Test type: Superiority or Other; Mean Difference (Final Values) = 1.12, 95% CI 2-sided [-0.81 to 3.04]
Statistical Analysis 35: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 33]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.66, 95% CI 2-sided [-1.26 to 2.57]
Statistical Analysis 36: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 33]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.34, 95% CI 2-sided [-1.57 to 2.25]
Statistical Analysis 37: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = 1.88, 95% CI 2-sided [-0.31 to 4.07]
Statistical Analysis 38: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.93, 95% CI 2-sided [-1.28 to 3.13]
Statistical Analysis 39: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.43, 95% CI 2-sided [-1.76 to 2.62]
Statistical Analysis 40: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.55, 95% CI 2-sided [-1.63 to 2.74]

10. Secondary Outcome: Change From Baseline in Swollen-Joint Counts at Week 12 (Descriptive Statistics)
Description: as for outcome 7
Time Frame: Week 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | PF-04171327 1 mg | PF-04171327 5 mg | PF-04171327 10 mg | PF-04171327 15 mg | Prednisone 5 mg | Prednisone 10 mg | Placebo
Number analyzed (Participants) | 44 | 41 | 44 | 43 | 44 | 43 | 41
Joints | -6.20 (6.21) | -5.98 (4.81) | -5.86 (6.17) | -5.58 (6.24) | -7.43 (5.82) | -7.07 (5.02) | -6.17 (5.48)

11. Secondary Outcome: Change From Baseline in C Reactive Protein (CRP) at Weeks 2, 4, 6, and 8 (Comparisons to Placebo and Prednisone 10 mg)
Description: The CRP was collected at each applicable clinic visit and analyzed by a central laboratory. In order to assist with the data clean-up at the end of the study, the CRP results were unblinded to the sponsor at the time of the last subject's last visit. All statistics presented below are derived from mixed model with fixed effects for treatment, visit, treatment-by-visit interaction and baseline value; unstructured covariance matrix was used.
Time Frame: Weeks 2, 4, 6, and 8
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | PF-04171327 1 mg | PF-04171327 5 mg | PF-04171327 10 mg | PF-04171327 15 mg | Prednisone 5 mg | Prednisone 10 mg | Placebo
Number analyzed (Participants) | 45 | 47 | 45 | 48 | 45 | 46 | 47
mg/L
  Week 2: number analyzed (Participants) | 44 | 46 | 45 | 48 | 45 | 45 | 44
  Week 2 | -7.29 (2.89) | -12.95 (2.82) | -13.73 (2.87) | -18.92 (2.78) | -8.25 (2.87) | -16.90 (2.86) | -2.80 (2.89)
  Week 4: number analyzed (Participants) | 45 | 43 | 43 | 44 | 43 | 45 | 45
  Week 4 | -9.77 (2.77) | -14.33 (2.78) | -11.52 (2.81) | -16.57 (2.75) | -3.92 (2.81) | -17.49 (2.76) | -6.35 (2.77)
  Week 6: number analyzed (Participants) | 44 | 43 | 45 | 44 | 44 | 46 | 43
  Week 6 | -9.35 (2.51) | -16.16 (2.53) | -13.05 (2.49) | -13.81 (2.51) | -6.54 (2.52) | -16.85 (2.46) | -3.93 (2.53)
  Week 8: number analyzed (Participants) | 43 | 42 | 44 | 43 | 43 | 45 | 43
  Week 8 | -7.29 (2.49) | -14.28 (2.52) | -14.86 (2.47) | -11.98 (2.49) | -7.23 (2.50) | -17.59 (2.44) | -4.19 (2.49)
Statistical Analysis 1: Comparison: PF-04171327 1 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -4.49, 95% CI 2-sided [-12.52 to 3.55]
Statistical Analysis 2: Comparison: PF-04171327 5 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -10.15, 95% CI 2-sided [-18.10 to -2.20]
Statistical Analysis 3: Comparison: PF-04171327 10 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -10.93, 95% CI 2-sided [-18.94 to -2.92]
Statistical Analysis 4: Comparison: PF-04171327 15 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -16.12, 95% CI 2-sided [-24.01 to -8.24]
Statistical Analysis 5: Comparison: Prednisone 5 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -5.45, 95% CI 2-sided [-13.45 to 2.56]
Statistical Analysis 6: Comparison: Prednisone 10 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -14.10, 95% CI 2-sided [-22.09 to -6.11]
Statistical Analysis 7: Comparison: PF-04171327 1 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -3.42, 95% CI 2-sided [-11.13 to 4.29]
Statistical Analysis 8: Comparison: PF-04171327 5 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -7.98, 95% CI 2-sided [-15.70 to -0.26]
Statistical Analysis 9: Comparison: PF-04171327 10 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -5.17, 95% CI 2-sided [-12.93 to 2.59]
Statistical Analysis 10: Comparison: PF-04171327 15 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -10.22, 95% CI 2-sided [-17.90 to -2.54]
Statistical Analysis 11: Comparison: Prednisone 5 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = 2.43, 95% CI 2-sided [-5.32 to 10.19]
Statistical Analysis 12: Comparison: Prednisone 10 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -11.14, 95% CI 2-sided [-18.83 to -3.45]
Statistical Analysis 13: Comparison: PF-04171327 1 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -5.42, 95% CI 2-sided [-12.44 to 1.59]
Statistical Analysis 14: Comparison: PF-04171327 5 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -12.24, 95% CI 2-sided [-19.27 to -5.20]
Statistical Analysis 15: Comparison: PF-04171327 10 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -9.13, 95% CI 2-sided [-16.11 to -2.14]
Statistical Analysis 16: Comparison: PF-04171327 15 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -9.88, 95% CI 2-sided [-16.89 to -2.88]
Statistical Analysis 17: Comparison: Prednisone 5 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -2.61, 95% CI 2-sided [-9.63 to 4.40]
Statistical Analysis 18: Comparison: Prednisone 10 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -12.93, 95% CI 2-sided [-19.88 to -5.98]
Statistical Analysis 19: Comparison: PF-04171327 1 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -3.10, 95% CI 2-sided [-10.03 to 3.83]
Statistical Analysis 20: Comparison: PF-04171327 5 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -10.10, 95% CI 2-sided [-17.06 to -3.13]
Statistical Analysis 21: Comparison: PF-04171327 10 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -10.67, 95% CI 2-sided [-17.57 to -3.77]
Statistical Analysis 22: Comparison: PF-04171327 15 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -7.79, 95% CI 2-sided [-14.72 to -0.86]
Statistical Analysis 23: Comparison: Prednisone 5 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -3.05, 95% CI 2-sided [-9.98 to 3.89]
Statistical Analysis 24: Comparison: Prednisone 10 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -13.41, 95% CI 2-sided [-20.27 to -6.54]
Statistical Analysis 25: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 25]; Test type: Superiority or Other; Mean Difference (Final Values) = 9.61, 95% CI 2-sided [1.62 to 17.61]
Statistical Analysis 26: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 25]; Test type: Superiority or Other; Mean Difference (Final Values) = 3.95, 95% CI 2-sided [-3.96 to 11.85]
Statistical Analysis 27: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 25]; Test type: Superiority or Other; Mean Difference (Final Values) = 3.17, 95% CI 2-sided [-4.80 to 11.13]
Statistical Analysis 28: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 25]; Test type: Superiority or Other; Mean Difference (Final Values) = -2.03, 95% CI 2-sided [-9.86 to 5.81]
Statistical Analysis 29: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = 7.72, 95% CI 2-sided [0.03 to 15.42]
Statistical Analysis 30: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = 3.16, 95% CI 2-sided [-4.54 to 10.87]
Statistical Analysis 31: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = 5.97, 95% CI 2-sided [-1.77 to 13.71]
Statistical Analysis 32: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.92, 95% CI 2-sided [-6.75 to 8.59]
Statistical Analysis 33: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 33]; Test type: Superiority or Other; Mean Difference (Final Values) = 7.50, 95% CI 2-sided [0.57 to 14.43]
Statistical Analysis 34: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 33]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.69, 95% CI 2-sided [-6.26 to 7.64]
Statistical Analysis 35: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 33]; Test type: Superiority or Other; Mean Difference (Final Values) = 3.80, 95% CI 2-sided [-3.09 to 10.70]
Statistical Analysis 36: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 33]; Test type: Superiority or Other; Mean Difference (Final Values) = 3.05, 95% CI 2-sided [-3.87 to 9.96]
Statistical Analysis 37: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = 10.31, 95% CI 2-sided [3.43 to 17.18]
Statistical Analysis 38: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = 3.31, 95% CI 2-sided [-3.59 to 10.22]
Statistical Analysis 39: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = 2.73, 95% CI 2-sided [-4.10 to 9.57]
Statistical Analysis 40: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = 5.62, 95% CI 2-sided [-1.25 to 12.48]

12. Secondary Outcome: Change From Baseline of CRP at Week 12 (Descriptive Statistics)
Description: The CRP was collected at each applicable clinic visit and analyzed by a central laboratory. In order to assist with the data clean-up at the end of the study, the CRP results were unblinded to the sponsor at the time of the last subject's last visit.
Time Frame: Week 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | PF-04171327 1 mg | PF-04171327 5 mg | PF-04171327 10 mg | PF-04171327 15 mg | Prednisone 5 mg | Prednisone 10 mg | Placebo
Number analyzed (Participants) | 42 | 39 | 43 | 42 | 43 | 42 | 39
mg/L | 0.72 (27.40) | -6.24 (23.06) | -4.52 (20.35) | -0.64 (29.08) | -2.90 (16.10) | -9.39 (36.10) | -4.07 (22.10)

13. Secondary Outcome: Change From Baseline in Patient Global Assessment of Arthritis at Weeks 2, 4, 6, and 8 (Comparisons to Placebo, and Prednisone 10 mg)
Description: Participants answered the following question, "Considering all the ways your arthritis affects you, how are you feeling today?" The subject's response was recorded using a 100 mm Visual Analog Scale (VAS), where 0 mm = no pain and 100 mm = most severe pain.
Time Frame: Weeks 2, 4, 6, and 8
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | PF-04171327 1 mg | PF-04171327 5 mg | PF-04171327 10 mg | PF-04171327 15 mg | Prednisone 5 mg | Prednisone 10 mg | Placebo
Number analyzed (Participants) | 45 | 47 | 45 | 48 | 45 | 46 | 47
mm
  Week 2: number analyzed (Participants) | 44 | 46 | 45 | 47 | 45 | 45 | 44
  Week 2 | -10.24 (2.85) | -18.77 (2.79) | -24.72 (2.83) | -22.50 (2.77) | -10.04 (2.83) | -23.51 (2.84) | -10.61 (2.85)
  Week 4: number analyzed (Participants) | 45 | 44 | 44 | 45 | 44 | 44 | 45
  Week 4 | -14.93 (3.21) | -24.04 (3.22) | -27.98 (3.24) | -23.14 (3.19) | -17.16 (3.24) | -28.31 (3.24) | -14.56 (3.21)
  Week 6: number analyzed (Participants) | 43 | 42 | 44 | 44 | 44 | 44 | 44
  Week 6 | -18.77 (3.28) | -30.84 (3.28) | -35.00 (3.27) | -27.93 (3.24) | -23.07 (3.27) | -32.34 (3.27) | -18.55 (3.26)
  Week 8: number analyzed (Participants) | 44 | 42 | 44 | 44 | 44 | 44 | 43
  Week 8 | -16.51 (3.49) | -29.08 (3.52) | -36.88 (3.50) | -31.32 (3.47) | -25.82 (3.50) | -34.60 (3.51) | -18.36 (3.51)
Statistical Analysis 1: Comparison: PF-04171327 1 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.38, 95% CI 2-sided [-7.56 to 8.31]
Statistical Analysis 2: Comparison: PF-04171327 5 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -8.15, 95% CI 2-sided [-16.01 to -0.30]
Statistical Analysis 3: Comparison: PF-04171327 10 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -14.10, 95% CI 2-sided [-22.01 to -6.20]
Statistical Analysis 4: Comparison: PF-04171327 15 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -11.88, 95% CI 2-sided [-19.70 to -4.06]
Statistical Analysis 5: Comparison: Prednisone 5 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.58, 95% CI 2-sided [-7.33 to 8.48]
Statistical Analysis 6: Comparison: Prednisone 10 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -12.89, 95% CI 2-sided [-20.80 to -4.98]
Statistical Analysis 7: Comparison: PF-04171327 1 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-9.31 to 8.58]
Statistical Analysis 8: Comparison: PF-04171327 5 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -9.48, 95% CI 2-sided [-18.43 to -0.53]
Statistical Analysis 9: Comparison: PF-04171327 10 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -13.42, 95% CI 2-sided [-22.39 to -4.44]
Statistical Analysis 10: Comparison: PF-04171327 15 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -8.58, 95% CI 2-sided [-17.48 to 0.33]
Statistical Analysis 11: Comparison: Prednisone 5 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -2.60, 95% CI 2-sided [-11.57 to 6.38]
Statistical Analysis 12: Comparison: Prednisone 10 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -13.75, 95% CI 2-sided [-22.73 to -4.78]
Statistical Analysis 13: Comparison: PF-04171327 1 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-9.32 to 8.88]
Statistical Analysis 14: Comparison: PF-04171327 5 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -12.28, 95% CI 2-sided [-21.39 to -3.17]
Statistical Analysis 15: Comparison: PF-04171327 10 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -16.44, 95% CI 2-sided [-25.53 to -7.36]
Statistical Analysis 16: Comparison: PF-04171327 15 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -9.38, 95% CI 2-sided [-18.42 to -0.34]
Statistical Analysis 17: Comparison: Prednisone 5 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -4.52, 95% CI 2-sided [-13.61 to 4.57]
Statistical Analysis 18: Comparison: Prednisone 10 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -13.78, 95% CI 2-sided [-22.87 to -4.69]
Statistical Analysis 19: Comparison: PF-04171327 1 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = 1.85, 95% CI 2-sided [-7.90 to 11.60]
Statistical Analysis 20: Comparison: PF-04171327 5 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -10.72, 95% CI 2-sided [-20.51 to -0.93]
Statistical Analysis 21: Comparison: PF-04171327 10 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -18.52, 95% CI 2-sided [-28.28 to -8.77]
Statistical Analysis 22: Comparison: PF-04171327 15 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -12.96, 95% CI 2-sided [-22.67 to -3.25]
Statistical Analysis 23: Comparison: Prednisone 5 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -7.46, 95% CI 2-sided [-17.21 to 2.30]
Statistical Analysis 24: Comparison: Prednisone 10 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -16.24, 95% CI 2-sided [-26.00 to -6.48]
Statistical Analysis 25: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 25]; Test type: Superiority or Other; Mean Difference (Final Values) = 13.27, 95% CI 2-sided [5.34 to 21.20]
Statistical Analysis 26: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 25]; Test type: Superiority or Other; Mean Difference (Final Values) = 4.74, 95% CI 2-sided [-3.12 to 12.59]
Statistical Analysis 27: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 25]; Test type: Superiority or Other; Mean Difference (Final Values) = -1.21, 95% CI 2-sided [-9.10 to 6.68]
Statistical Analysis 28: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 25]; Test type: Superiority or Other; Mean Difference (Final Values) = 1.01, 95% CI 2-sided [-6.79 to 8.81]
Statistical Analysis 29: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = 13.39, 95% CI 2-sided [4.39 to 22.38]
Statistical Analysis 30: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = 4.27, 95% CI 2-sided [-4.73 to 13.27]
Statistical Analysis 31: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.34, 95% CI 2-sided [-8.68 to 9.35]
Statistical Analysis 32: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = 5.18, 95% CI 2-sided [-3.77 to 14.12]
Statistical Analysis 33: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 33]; Test type: Superiority or Other; Mean Difference (Final Values) = 13.56, 95% CI 2-sided [4.44 to 22.68]
Statistical Analysis 34: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 33]; Test type: Superiority or Other; Mean Difference (Final Values) = 1.50, 95% CI 2-sided [-7.64 to 10.64]
Statistical Analysis 35: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 33]; Test type: Superiority or Other; Mean Difference (Final Values) = -2.66, 95% CI 2-sided [-11.76 to 6.44]
Statistical Analysis 36: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 33]; Test type: Superiority or Other; Mean Difference (Final Values) = 4.41, 95% CI 2-sided [-4.65 to 13.46]
Statistical Analysis 37: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = 18.09, 95% CI 2-sided [8.34 to 27.84]
Statistical Analysis 38: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = 5.52, 95% CI 2-sided [-4.27 to 15.32]
Statistical Analysis 39: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = -2.28, 95% CI 2-sided [-12.03 to 7.46]
Statistical Analysis 40: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = 3.28, 95% CI 2-sided [-6.42 to 12.98]

14. Secondary Outcome: Change From Baseline in Patient Global Assessment of Arthritis at Week 12 (Descriptive Statistics)
Description: as for outcome 13
Time Frame: Week 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | PF-04171327 1 mg | PF-04171327 5 mg | PF-04171327 10 mg | PF-04171327 15 mg | Prednisone 5 mg | Prednisone 10 mg | Placebo
Number analyzed (Participants) | 44 | 41 | 44 | 43 | 44 | 42 | 41
mm | -14.54 (27.33) | -22.26 (26.11) | -18.10 (25.35) | -16.74 (31.57) | -19.24 (29.32) | -25.29 (29.20) | -17.90 (23.14)

15. Secondary Outcome: Change From Baseline in Physician Global Assessment of Arthritis at Weeks 2, 4, 6, and 8 (Comparisons to Placebo, and Prednisone 10 mg)
Description: The investigator assessed how the participant's overall arthritis appears at the time of the visit. This was an evaluation based on the participant's disease signs, functional capacity and physical examination, and was independent of the Patient's Global Assessment of Arthritis. The investigator's response was recorded using a 100 mm VAS, where 0 mm = no pain and 100 mm = most severe pain.
Time Frame: Weeks 2, 4, 6, and 8
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | PF-04171327 1 mg | PF-04171327 5 mg | PF-04171327 10 mg | PF-04171327 15 mg | Prednisone 5 mg | Prednisone 10 mg | Placebo
Number analyzed (Participants) | 45 | 47 | 45 | 48 | 45 | 46 | 47
mm
  Week 2: number analyzed (Participants) | 43 | 46 | 45 | 47 | 45 | 45 | 44
  Week 2 | -16.35 (2.53) | -21.74 (2.45) | -22.14 (2.48) | -25.21 (2.43) | -13.24 (2.48) | -22.80 (2.48) | -9.29 (2.50)
  Week 4: number analyzed (Participants) | 43 | 44 | 44 | 45 | 44 | 44 | 45
  Week 4 | -22.25 (2.68) | -27.03 (2.64) | -30.72 (2.66) | -28.95 (2.62) | -20.94 (2.66) | -31.16 (2.66) | -15.00 (2.64)
  Week 6: number analyzed (Participants) | 43 | 42 | 44 | 44 | 44 | 44 | 44
  Week 6 | -25.58 (2.68) | -32.54 (2.67) | -34.79 (2.66) | -32.79 (2.63) | -28.54 (2.66) | -33.92 (2.66) | -19.48 (2.65)
  Week 8: number analyzed (Participants) | 43 | 42 | 44 | 44 | 44 | 44 | 43
  Week 8 | -26.24 (2.81) | -33.92 (2.82) | -38.00 (2.79) | -33.71 (2.77) | -29.25 (2.79) | -35.50 (2.79) | -21.52 (2.79)
Statistical Analysis 1: Comparison: PF-04171327 1 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -7.06, 95% CI 2-sided [-14.07 to -0.06]
Statistical Analysis 2: Comparison: PF-04171327 5 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -12.45, 95% CI 2-sided [-19.34 to -5.56]
Statistical Analysis 3: Comparison: PF-04171327 10 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -12.85, 95% CI 2-sided [-19.79 to -5.91]
Statistical Analysis 4: Comparison: PF-04171327 15 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -15.92, 95% CI 2-sided [-22.79 to -9.06]
Statistical Analysis 5: Comparison: Prednisone 5 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -3.95, 95% CI 2-sided [-10.89 to 2.99]
Statistical Analysis 6: Comparison: Prednisone 10 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -13.51, 95% CI 2-sided [-20.44 to -6.57]
Statistical Analysis 7: Comparison: PF-04171327 1 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -7.25, 95% CI 2-sided [-14.65 to 0.16]
Statistical Analysis 8: Comparison: PF-04171327 5 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -12.03, 95% CI 2-sided [-19.38 to -4.68]
Statistical Analysis 9: Comparison: PF-04171327 10 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -15.72, 95% CI 2-sided [-23.10 to -8.35]
Statistical Analysis 10: Comparison: PF-04171327 15 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -13.95, 95% CI 2-sided [-21.27 to -6.63]
Statistical Analysis 11: Comparison: Prednisone 5 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -5.94, 95% CI 2-sided [-13.31 to 1.43]
Statistical Analysis 12: Comparison: Prednisone 10 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -16.16, 95% CI 2-sided [-23.54 to -8.79]
Statistical Analysis 13: Comparison: PF-04171327 1 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -6.09, 95% CI 2-sided [-13.50 to 1.32]
Statistical Analysis 14: Comparison: PF-04171327 5 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -13.06, 95% CI 2-sided [-20.46 to -5.65]
Statistical Analysis 15: Comparison: PF-04171327 10 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -15.31, 95% CI 2-sided [-22.69 to -7.93]
Statistical Analysis 16: Comparison: PF-04171327 15 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -13.31, 95% CI 2-sided [-20.66 to -5.96]
Statistical Analysis 17: Comparison: Prednisone 5 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -9.06, 95% CI 2-sided [-16.44 to -1.68]
Statistical Analysis 18: Comparison: Prednisone 10 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -14.44, 95% CI 2-sided [-21.82 to -7.06]
Statistical Analysis 19: Comparison: PF-04171327 1 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -4.72, 95% CI 2-sided [-12.53 to 3.09]
Statistical Analysis 20: Comparison: PF-04171327 5 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -12.40, 95% CI 2-sided [-20.21 to -4.59]
Statistical Analysis 21: Comparison: PF-04171327 10 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -16.48, 95% CI 2-sided [-24.25 to -8.71]
Statistical Analysis 22: Comparison: PF-04171327 15 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -12.19, 95% CI 2-sided [-19.94 to -4.44]
Statistical Analysis 23: Comparison: Prednisone 5 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -7.73, 95% CI 2-sided [-15.50 to 0.04]
Statistical Analysis 24: Comparison: Prednisone 10 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -13.98, 95% CI 2-sided [-21.75 to -6.21]
Statistical Analysis 25: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 25]; Test type: Superiority or Other; Mean Difference (Final Values) = 6.45, 95% CI 2-sided [-0.53 to 13.42]
Statistical Analysis 26: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 25]; Test type: Superiority or Other; Mean Difference (Final Values) = 1.06, 95% CI 2-sided [-5.81 to 7.92]
Statistical Analysis 27: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 25]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.66, 95% CI 2-sided [-6.25 to 7.57]
Statistical Analysis 28: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 25]; Test type: Superiority or Other; Mean Difference (Final Values) = -2.42, 95% CI 2-sided [-9.26 to 4.42]
Statistical Analysis 29: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = 8.91, 95% CI 2-sided [1.48 to 16.35]
Statistical Analysis 30: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = 4.13, 95% CI 2-sided [-3.24 to 11.51]
Statistical Analysis 31: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.44, 95% CI 2-sided [-6.96 to 7.84]
Statistical Analysis 32: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = 2.21, 95% CI 2-sided [-5.14 to 9.56]
Statistical Analysis 33: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 33]; Test type: Superiority or Other; Mean Difference (Final Values) = 8.35, 95% CI 2-sided [0.92 to 15.77]
Statistical Analysis 34: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 33]; Test type: Superiority or Other; Mean Difference (Final Values) = 1.38, 95% CI 2-sided [-6.03 to 8.80]
Statistical Analysis 35: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 33]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.87, 95% CI 2-sided [-8.26 to 6.52]
Statistical Analysis 36: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 33]; Test type: Superiority or Other; Mean Difference (Final Values) = 1.13, 95% CI 2-sided [-6.23 to 8.49]
Statistical Analysis 37: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = 9.26, 95% CI 2-sided [1.46 to 17.06]
Statistical Analysis 38: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = 1.58, 95% CI 2-sided [-6.23 to 9.38]
Statistical Analysis 39: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = -2.50, 95% CI 2-sided [-10.27 to 5.27]
Statistical Analysis 40: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = 1.79, 95% CI 2-sided [-5.95 to 9.53]

16. Secondary Outcome: Change From Baseline in Physician Global Assessment of Arthritis at Week 12 (Descriptive Statistics)
Description: as for outcome 15
Time Frame: Week 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | PF-04171327 1 mg | PF-04171327 5 mg | PF-04171327 10 mg | PF-04171327 15 mg | Prednisone 5 mg | Prednisone 10 mg | Placebo
Number analyzed (Participants) | 43 | 41 | 44 | 43 | 44 | 42 | 40
mm | -25.00 (21.57) | -28.56 (26.41) | -23.04 (22.00) | -24.30 (28.15) | -27.25 (23.71) | -27.25 (20.42) | -19.34 (27.21)

17. Secondary Outcome: Change From Baseline in Pain VAS at Weeks 2, 4, 6, and 8 (Comparisons to Placebo, and Prednisone 10 mg)
Description: Participants assessed the severity of their arthritis pain using a 100 mm VAS placing a mark on the scale between 0 (no pain) and 100 (most severe pain), which corresponds to the magnitude of their pain.
Time Frame: Weeks 2, 4, 6, and 8
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | PF-04171327 1 mg | PF-04171327 5 mg | PF-04171327 10 mg | PF-04171327 15 mg | Prednisone 5 mg | Prednisone 10 mg | Placebo
Number analyzed (Participants) | 45 | 47 | 45 | 48 | 45 | 46 | 47
mm
  Week 2: number analyzed (Participants) | 44 | 46 | 45 | 47 | 45 | 45 | 44
  Week 2 | -13.41 (2.88) | -17.40 (2.83) | -24.90 (2.86) | -22.86 (2.80) | -12.68 (2.86) | -24.59 (2.87) | -10.54 (2.88)
  Week 4: number analyzed (Participants) | 45 | 44 | 44 | 45 | 44 | 44 | 45
  Week 4 | -15.55 (3.08) | -24.38 (3.09) | -29.70 (3.10) | -26.08 (3.05) | -20.26 (3.10) | -29.65 (3.11) | -14.28 (3.08)
  Week 6: number analyzed (Participants) | 43 | 42 | 44 | 44 | 44 | 44 | 44
  Week 6 | -19.03 (3.33) | -29.16 (3.35) | -34.37 (3.33) | -30.15 (3.30) | -24.16 (3.33) | -34.69 (3.34) | -18.80 (3.32)
  Week 8: number analyzed (Participants) | 44 | 42 | 44 | 44 | 44 | 44 | 43
  Week 8 | -18.95 (3.45) | -28.53 (3.50) | -37.96 (3.46) | -30.91 (3.43) | -25.86 (3.46) | -37.60 (3.47) | -18.26 (3.47)
Statistical Analysis 1: Comparison: PF-04171327 1 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -2.87, 95% CI 2-sided [-10.89 to 5.14]
Statistical Analysis 2: Comparison: PF-04171327 5 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -6.86, 95% CI 2-sided [-14.80 to 1.08]
Statistical Analysis 3: Comparison: PF-04171327 10 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -14.36, 95% CI 2-sided [-22.34 to -6.38]
Statistical Analysis 4: Comparison: PF-04171327 15 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -12.32, 95% CI 2-sided [-20.22 to -4.41]
Statistical Analysis 5: Comparison: Prednisone 5 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -2.14, 95% CI 2-sided [-10.12 to 5.85]
Statistical Analysis 6: Comparison: Prednisone 10 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -14.05, 95% CI 2-sided [-22.05 to -6.04]
Statistical Analysis 7: Comparison: PF-04171327 1 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -1.26, 95% CI 2-sided [-9.83 to 7.30]
Statistical Analysis 8: Comparison: PF-04171327 5 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -10.10, 95% CI 2-sided [-18.67 to -1.53]
Statistical Analysis 9: Comparison: PF-04171327 10 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -15.41, 95% CI 2-sided [-24.01 to -6.82]
Statistical Analysis 10: Comparison: PF-04171327 15 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -11.79, 95% CI 2-sided [-20.33 to -3.26]
Statistical Analysis 11: Comparison: Prednisone 5 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -5.98, 95% CI 2-sided [-14.57 to 2.62]
Statistical Analysis 12: Comparison: Prednisone 10 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -15.37, 95% CI 2-sided [-23.98 to -6.76]
Statistical Analysis 13: Comparison: PF-04171327 1 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-9.49 to 9.03]
Statistical Analysis 14: Comparison: PF-04171327 5 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -10.36, 95% CI 2-sided [-19.64 to -1.08]
Statistical Analysis 15: Comparison: PF-04171327 10 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -15.57, 95% CI 2-sided [-24.83 to -6.32]
Statistical Analysis 16: Comparison: PF-04171327 15 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -11.34, 95% CI 2-sided [-20.56 to -2.13]
Statistical Analysis 17: Comparison: Prednisone 5 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -5.36, 95% CI 2-sided [-14.61 to 3.89]
Statistical Analysis 18: Comparison: Prednisone 10 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -15.88, 95% CI 2-sided [-25.15 to -6.61]
Statistical Analysis 19: Comparison: PF-04171327 1 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.69, 95% CI 2-sided [-10.32 to 8.94]
Statistical Analysis 20: Comparison: PF-04171327 5 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -10.27, 95% CI 2-sided [-19.95 to -0.59]
Statistical Analysis 21: Comparison: PF-04171327 10 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -19.70, 95% CI 2-sided [-29.34 to -10.06]
Statistical Analysis 22: Comparison: PF-04171327 15 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -12.65, 95% CI 2-sided [-22.25 to -3.04]
Statistical Analysis 23: Comparison: Prednisone 5 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -7.60, 95% CI 2-sided [-17.24 to 2.04]
Statistical Analysis 24: Comparison: Prednisone 10 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -19.34, 95% CI 2-sided [-28.99 to -9.68]
Statistical Analysis 25: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 25]; Test type: Superiority or Other; Mean Difference (Final Values) = 11.17, 95% CI 2-sided [3.18 to 19.16]
Statistical Analysis 26: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 25]; Test type: Superiority or Other; Mean Difference (Final Values) = 7.19, 95% CI 2-sided [-0.78 to 15.15]
Statistical Analysis 27: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 25]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.31, 95% CI 2-sided [-8.28 to 7.65]
Statistical Analysis 28: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 25]; Test type: Superiority or Other; Mean Difference (Final Values) = 1.73, 95% CI 2-sided [-6.14 to 9.61]
Statistical Analysis 29: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = 14.11, 95% CI 2-sided [5.51 to 22.71]
Statistical Analysis 30: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = 5.27, 95% CI 2-sided [-3.38 to 13.92]
Statistical Analysis 31: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-8.68 to 8.59]
Statistical Analysis 32: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = 3.58, 95% CI 2-sided [-4.99 to 12.15]
Statistical Analysis 33: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 33]; Test type: Superiority or Other; Mean Difference (Final Values) = 15.65, 95% CI 2-sided [6.38 to 24.93]
Statistical Analysis 34: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 33]; Test type: Superiority or Other; Mean Difference (Final Values) = 5.53, 95% CI 2-sided [-3.81 to 14.86]
Statistical Analysis 35: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 33]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.31, 95% CI 2-sided [-8.97 to 9.59]
Statistical Analysis 36: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 33]; Test type: Superiority or Other; Mean Difference (Final Values) = 4.54, 95% CI 2-sided [-4.69 to 13.77]
Statistical Analysis 37: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = 18.65, 95% CI 2-sided [9.03 to 28.27]
Statistical Analysis 38: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = 9.07, 95% CI 2-sided [-0.64 to 18.78]
Statistical Analysis 39: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-10.00 to 9.28]
Statistical Analysis 40: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = 6.69, 95% CI 2-sided [-2.91 to 16.29]

18. Secondary Outcome: Change From Baseline in Pain VAS at Week 12 (Descriptive Statistics)
Description: as for outcome 17
Time Frame: Week 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | PF-04171327 1 mg | PF-04171327 5 mg | PF-04171327 10 mg | PF-04171327 15 mg | Prednisone 5 mg | Prednisone 10 mg | Placebo
Number analyzed (Participants) | 44 | 40 | 44 | 43 | 44 | 42 | 41
mm | -17.86 (26.70) | -19.40 (29.04) | -18.23 (27.75) | -16.60 (30.50) | -21.52 (24.69) | -25.17 (29.60) | -16.30 (22.41)

19. Secondary Outcome: Change From Baseline in HAQ-DI at Weeks 2, 4, 6, and 8 (Comparisons to Placebo, and Prednisone 10 mg)
Description: Health Assessment Questionnaire-Disability Index (HAQ-DI): participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: Weeks 2, 4, 6, and 8
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | PF-04171327 1 mg | PF-04171327 5 mg | PF-04171327 10 mg | PF-04171327 15 mg | Prednisone 5 mg | Prednisone 10 mg | Placebo
Number analyzed (Participants) | 45 | 47 | 45 | 48 | 45 | 46 | 47
Units on a scale
  Week 2: number analyzed (Participants) | 44 | 46 | 45 | 47 | 45 | 45 | 44
  Week 2 | -0.25 (0.06) | -0.34 (0.06) | -0.33 (0.06) | -0.41 (0.06) | -0.23 (0.06) | -0.41 (0.06) | -0.05 (0.06)
  Week 4: number analyzed (Participants) | 45 | 44 | 44 | 45 | 44 | 44 | 45
  Week 4 | -0.26 (0.07) | -0.50 (0.07) | -0.43 (0.07) | -0.51 (0.07) | -0.34 (0.07) | -0.58 (0.07) | -0.14 (0.07)
  Week 6: number analyzed (Participants) | 44 | 42 | 44 | 44 | 44 | 44 | 44
  Week 6 | -0.35 (0.07) | -0.60 (0.07) | -0.52 (0.07) | -0.56 (0.07) | -0.39 (0.07) | -0.68 (0.07) | -0.21 (0.07)
  Week 8: number analyzed (Participants) | 44 | 42 | 44 | 44 | 44 | 44 | 43
  Week 8 | -0.26 (0.08) | -0.59 (0.08) | -0.60 (0.08) | -0.55 (0.08) | -0.50 (0.08) | -0.77 (0.08) | -0.19 (0.08)
Statistical Analysis 1: Comparison: PF-04171327 1 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.37 to -0.02]
Statistical Analysis 2: Comparison: PF-04171327 5 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.29, 95% CI 2-sided [-0.46 to -0.11]
Statistical Analysis 3: Comparison: PF-04171327 10 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-0.45 to -0.10]
Statistical Analysis 4: Comparison: PF-04171327 15 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-0.52 to -0.18]
Statistical Analysis 5: Comparison: Prednisone 5 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.35 to 0.00]
Statistical Analysis 6: Comparison: Prednisone 10 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-0.53 to -0.18]
Statistical Analysis 7: Comparison: PF-04171327 1 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.31 to 0.07]
Statistical Analysis 8: Comparison: PF-04171327 5 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-0.54 to -0.17]
Statistical Analysis 9: Comparison: PF-04171327 10 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-0.47 to -0.09]
Statistical Analysis 10: Comparison: PF-04171327 15 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-0.56 to -0.18]
Statistical Analysis 11: Comparison: Prednisone 5 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-0.39 to -0.01]
Statistical Analysis 12: Comparison: Prednisone 10 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-0.63 to -0.25]
Statistical Analysis 13: Comparison: PF-04171327 1 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.34 to 0.05]
Statistical Analysis 14: Comparison: PF-04171327 5 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-0.59 to -0.20]
Statistical Analysis 15: Comparison: PF-04171327 10 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.32, 95% CI 2-sided [-0.51 to -0.12]
Statistical Analysis 16: Comparison: PF-04171327 15 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-0.55 to -0.16]
Statistical Analysis 17: Comparison: Prednisone 5 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.38 to 0.01]
Statistical Analysis 18: Comparison: Prednisone 10 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-0.67 to -0.27]
Statistical Analysis 19: Comparison: PF-04171327 1 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.30 to 0.15]
Statistical Analysis 20: Comparison: PF-04171327 5 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-0.63 to -0.18]
Statistical Analysis 21: Comparison: PF-04171327 10 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.41, 95% CI 2-sided [-0.64 to -0.18]
Statistical Analysis 22: Comparison: PF-04171327 15 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-0.59 to -0.14]
Statistical Analysis 23: Comparison: Prednisone 5 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.32, 95% CI 2-sided [-0.54 to -0.09]
Statistical Analysis 24: Comparison: Prednisone 10 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.58, 95% CI 2-sided [-0.81 to -0.35]
Statistical Analysis 25: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 25]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.16, 95% CI 2-sided [-0.01 to 0.34]
Statistical Analysis 26: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 25]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.10 to 0.24]
Statistical Analysis 27: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 25]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-0.10 to 0.25]
Statistical Analysis 28: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 25]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.17 to 0.18]
Statistical Analysis 29: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.32, 95% CI 2-sided [0.13 to 0.51]
Statistical Analysis 30: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-0.11 to 0.27]
Statistical Analysis 31: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [-0.04 to 0.34]
Statistical Analysis 32: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.13 to 0.25]
Statistical Analysis 33: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 33]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.32, 95% CI 2-sided [0.13 to 0.52]
Statistical Analysis 34: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 33]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.12 to 0.27]
Statistical Analysis 35: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 33]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [-0.05 to 0.35]
Statistical Analysis 36: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 33]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.08 to 0.31]
Statistical Analysis 37: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.51, 95% CI 2-sided [0.28 to 0.73]
Statistical Analysis 38: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [-0.05 to 0.40]
Statistical Analysis 39: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [-0.06 to 0.40]
Statistical Analysis 40: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.22, 95% CI 2-sided [-0.01 to 0.44]

20. Secondary Outcome: Change From Baseline in HAQ-DI at Week 12 (Descriptive Statistics)
Description: as for outcome 19
Time Frame: Week 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | PF-04171327 1 mg | PF-04171327 5 mg | PF-04171327 10 mg | PF-04171327 15 mg | Prednisone 5 mg | Prednisone 10 mg | Placebo
Number analyzed (Participants) | 44 | 41 | 44 | 43 | 44 | 42 | 41
Units on a scale | -0.28 (0.63) | -0.57 (0.65) | -0.37 (0.50) | -0.38 (0.50) | -0.52 (0.63) | -0.56 (0.59) | -0.26 (0.56)

21. Secondary Outcome: Change From Baseline in Disease Activity Score (DAS) 28-3 CRP at Weeks 2, 4, 6, and 8 (Comparisons to Placebo, and Prednisone 10 mg)
Description: DAS28-3 (CRP) was calculated from the SJC and TJC using the 28 joints count and CRP (mg/L). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-3 (CRP) <= 3.2 implied low disease activity and >3.2 to 5.1 implied moderate to high disease activity, and DAS28-3 (CRP) <2.6 = remission.
Time Frame: Weeks 2, 4, 6, and 8
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | PF-04171327 1 mg | PF-04171327 5 mg | PF-04171327 10 mg | PF-04171327 15 mg | Prednisone 5 mg | Prednisone 10 mg | Placebo
Number analyzed (Participants) | 45 | 47 | 45 | 48 | 45 | 46 | 47
Units on a scale
  Week 2: number analyzed (Participants) | 44 | 46 | 45 | 46 | 45 | 45 | 44
  Week 2 | -0.81 (0.13) | -1.15 (0.13) | -1.21 (0.13) | -1.51 (0.13) | -0.75 (0.13) | -1.23 (0.13) | -0.40 (0.13)
  Week 4: number analyzed (Participants) | 44 | 43 | 43 | 43 | 43 | 44 | 45
  Week 4 | -1.19 (0.15) | -1.49 (0.15) | -1.71 (0.15) | -1.73 (0.15) | -1.01 (0.15) | -1.67 (0.15) | -0.76 (0.15)
  Week 6: number analyzed (Participants) | 44 | 42 | 44 | 43 | 44 | 45 | 43
  Week 6 | -1.38 (0.16) | -1.81 (0.16) | -2.01 (0.16) | -1.99 (0.16) | -1.37 (0.16) | -1.98 (0.16) | -0.94 (0.16)
  Week 8: number analyzed (Participants) | 43 | 42 | 44 | 42 | 43 | 45 | 42
  Week 8 | -1.44 (0.17) | -1.84 (0.17) | -2.22 (0.17) | -2.13 (0.17) | -1.42 (0.17) | -2.14 (0.17) | -0.93 (0.17)
Statistical Analysis 1: Comparison: PF-04171327 1 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.41, 95% CI 2-sided [-0.78 to -0.04]
Statistical Analysis 2: Comparison: PF-04171327 5 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.75, 95% CI 2-sided [-1.12 to -0.39]
Statistical Analysis 3: Comparison: PF-04171327 10 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.81, 95% CI 2-sided [-1.18 to -0.44]
Statistical Analysis 4: Comparison: PF-04171327 15 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -1.11, 95% CI 2-sided [-1.48 to -0.74]
Statistical Analysis 5: Comparison: Prednisone 5 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-0.72 to 0.02]
Statistical Analysis 6: Comparison: Prednisone 10 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.83, 95% CI 2-sided [-1.19 to -0.46]
Statistical Analysis 7: Comparison: PF-04171327 1 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.43, 95% CI 2-sided [-0.85 to -0.00]
Statistical Analysis 8: Comparison: PF-04171327 5 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.73, 95% CI 2-sided [-1.15 to -0.31]
Statistical Analysis 9: Comparison: PF-04171327 10 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.95, 95% CI 2-sided [-1.37 to -0.52]
Statistical Analysis 10: Comparison: PF-04171327 15 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.96, 95% CI 2-sided [-1.39 to -0.54]
Statistical Analysis 11: Comparison: Prednisone 5 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.67 to 0.18]
Statistical Analysis 12: Comparison: Prednisone 10 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.91, 95% CI 2-sided [-1.33 to -0.49]
Statistical Analysis 13: Comparison: PF-04171327 1 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-0.90 to 0.02]
Statistical Analysis 14: Comparison: PF-04171327 5 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.87, 95% CI 2-sided [-1.32 to -0.41]
Statistical Analysis 15: Comparison: PF-04171327 10 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -1.07, 95% CI 2-sided [-1.53 to -0.62]
Statistical Analysis 16: Comparison: PF-04171327 15 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -1.05, 95% CI 2-sided [-1.51 to -0.60]
Statistical Analysis 17: Comparison: Prednisone 5 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.43, 95% CI 2-sided [-0.89 to 0.03]
Statistical Analysis 18: Comparison: Prednisone 10 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -1.04, 95% CI 2-sided [-1.50 to -0.59]
Statistical Analysis 19: Comparison: PF-04171327 1 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.51, 95% CI 2-sided [-1.00 to -0.03]
Statistical Analysis 20: Comparison: PF-04171327 5 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.91, 95% CI 2-sided [-1.40 to -0.43]
Statistical Analysis 21: Comparison: PF-04171327 10 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -1.29, 95% CI 2-sided [-1.77 to -0.80]
Statistical Analysis 22: Comparison: PF-04171327 15 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -1.20, 95% CI 2-sided [-1.69 to -0.72]
Statistical Analysis 23: Comparison: Prednisone 5 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.49, 95% CI 2-sided [-0.98 to -0.01]
Statistical Analysis 24: Comparison: Prednisone 10 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -1.21, 95% CI 2-sided [-1.69 to -0.73]
Statistical Analysis 25: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 25]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.41, 95% CI 2-sided [0.04 to 0.78]
Statistical Analysis 26: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 25]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.29 to 0.44]
Statistical Analysis 27: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 25]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.35 to 0.38]
Statistical Analysis 28: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 25]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.29, 95% CI 2-sided [-0.65 to 0.08]
Statistical Analysis 29: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.48, 95% CI 2-sided [0.06 to 0.91]
Statistical Analysis 30: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [-0.24 to 0.60]
Statistical Analysis 31: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.46 to 0.38]
Statistical Analysis 32: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.48 to 0.37]
Statistical Analysis 33: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 33]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.61, 95% CI 2-sided [0.15 to 1.06]
Statistical Analysis 34: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 33]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [-0.28 to 0.63]
Statistical Analysis 35: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 33]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.49 to 0.42]
Statistical Analysis 36: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 33]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.47 to 0.44]
Statistical Analysis 37: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.70, 95% CI 2-sided [0.22 to 1.18]
Statistical Analysis 38: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.30, 95% CI 2-sided [-0.18 to 0.78]
Statistical Analysis 39: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.55 to 0.40]
Statistical Analysis 40: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.47 to 0.49]

22. Secondary Outcome: Change From Baseline in DAS 28-3 CRP at Week 12 (Descriptive Statistics)
Description: as for outcome 21
Time Frame: Week 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | PF-04171327 1 mg | PF-04171327 5 mg | PF-04171327 10 mg | PF-04171327 15 mg | Prednisone 5 mg | Prednisone 10 mg | Placebo
Number analyzed (Participants) | 43 | 41 | 44 | 41 | 44 | 43 | 40
Units on a scale | -1.30 (1.21) | -1.37 (1.05) | -1.29 (1.14) | -1.25 (1.36) | -1.45 (1.05) | -1.62 (1.00) | -1.13 (1.08)

23. Secondary Outcome: Change From Baseline in DAS28-4(CRP) at Weeks 2, 4, 6, and 8 (Comparisons to Placebo, and Prednisone 10 mg)
Description: DAS28-4 (CRP) was calculated from the SJC and TJC using the 28 joints count and CRP (mg/L). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-3 (CRP) <= 3.2 implied low disease activity and >3.2 to 5.1 implied moderate to high disease activity, and DAS28-3 (CRP) <2.6 = remission. All statistics presented below are derived from mixed model with fixed effects for treatment, visit, treatment-by-visit interaction and baseline value; unstructured covariance matrix was used.
Time Frame: Weeks 2, 4, 6, and 8
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | PF-04171327 1 mg | PF-04171327 5 mg | PF-04171327 10 mg | PF-04171327 15 mg | Prednisone 5 mg | Prednisone 10 mg | Placebo
Number analyzed (Participants) | 45 | 47 | 45 | 48 | 45 | 46 | 47
Units on a scale
  Week 2: number analyzed (Participants) | 44 | 46 | 45 | 46 | 45 | 44 | 44
  Week 2 | -0.88 (0.14) | -1.29 (0.14) | -1.45 (0.14) | -1.69 (0.14) | -0.82 (0.14) | -1.46 (0.14) | -0.52 (0.14)
  Week 4: number analyzed (Participants) | 44 | 43 | 43 | 43 | 43 | 43 | 45
  Week 4 | -1.29 (0.16) | -1.68 (0.16) | -1.97 (0.16) | -1.90 (0.16) | -1.15 (0.16) | -1.92 (0.16) | -0.90 (0.16)
  Week 6: number analyzed (Participants) | 44 | 42 | 44 | 43 | 44 | 44 | 43
  Week 6 | -1.51 (0.18) | -2.06 (0.18) | -2.32 (0.18) | -2.21 (0.18) | -1.56 (0.18) | -2.27 (0.18) | -1.12 (0.18)
  Week 8: number analyzed (Participants) | 43 | 42 | 44 | 42 | 43 | 44 | 42
  Week 8 | -1.55 (0.19) | -2.07 (0.19) | -2.53 (0.19) | -2.38 (0.19) | -1.65 (0.19) | -2.44 (0.19) | -1.11 (0.19)
Statistical Analysis 1: Comparison: PF-04171327 1 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-0.76 to 0.03]
Statistical Analysis 2: Comparison: PF-04171327 5 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.78, 95% CI 2-sided [-1.17 to -0.39]
Statistical Analysis 3: Comparison: PF-04171327 10 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.93, 95% CI 2-sided [-1.32 to -0.54]
Statistical Analysis 4: Comparison: PF-04171327 15 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -1.17, 95% CI 2-sided [-1.56 to -0.78]
Statistical Analysis 5: Comparison: Prednisone 5 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-0.70 to 0.09]
Statistical Analysis 6: Comparison: Prednisone 10 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.95, 95% CI 2-sided [-1.34 to -0.55]
Statistical Analysis 7: Comparison: PF-04171327 1 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-0.84 to 0.07]
Statistical Analysis 8: Comparison: PF-04171327 5 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.78, 95% CI 2-sided [-1.23 to -0.32]
Statistical Analysis 9: Comparison: PF-04171327 10 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -1.06, 95% CI 2-sided [-1.52 to -0.61]
Statistical Analysis 10: Comparison: PF-04171327 15 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -1.00, 95% CI 2-sided [-1.45 to -0.54]
Statistical Analysis 11: Comparison: Prednisone 5 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-0.71 to 0.21]
Statistical Analysis 12: Comparison: Prednisone 10 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -1.02, 95% CI 2-sided [-1.48 to -0.57]
Statistical Analysis 13: Comparison: PF-04171327 1 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-0.89 to 0.11]
Statistical Analysis 14: Comparison: PF-04171327 5 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.94, 95% CI 2-sided [-1.44 to -0.45]
Statistical Analysis 15: Comparison: PF-04171327 10 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -1.21, 95% CI 2-sided [-1.71 to -0.71]
Statistical Analysis 16: Comparison: PF-04171327 15 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -1.09, 95% CI 2-sided [-1.59 to -0.59]
Statistical Analysis 17: Comparison: Prednisone 5 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.45, 95% CI 2-sided [-0.95 to 0.05]
Statistical Analysis 18: Comparison: Prednisone 10 mg vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; Mean Difference (Final Values) = -1.15, 95% CI 2-sided [-1.65 to -0.66]
Statistical Analysis 19: Comparison: PF-04171327 1 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-0.96 to 0.08]
Statistical Analysis 20: Comparison: PF-04171327 5 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.96, 95% CI 2-sided [-1.48 to -0.44]
Statistical Analysis 21: Comparison: PF-04171327 10 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -1.43, 95% CI 2-sided [-1.94 to -0.91]
Statistical Analysis 22: Comparison: PF-04171327 15 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -1.28, 95% CI 2-sided [-1.80 to -0.76]
Statistical Analysis 23: Comparison: Prednisone 5 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.55, 95% CI 2-sided [-1.06 to -0.03]
Statistical Analysis 24: Comparison: Prednisone 10 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -1.33, 95% CI 2-sided [-1.85 to -0.81]
Statistical Analysis 25: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 25]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.59, 95% CI 2-sided [0.19 to 0.98]
Statistical Analysis 26: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 25]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [-0.22 to 0.56]
Statistical Analysis 27: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 25]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.38 to 0.41]
Statistical Analysis 28: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 25]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.62 to 0.16]
Statistical Analysis 29: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.64, 95% CI 2-sided [0.18 to 1.09]
Statistical Analysis 30: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.24, 95% CI 2-sided [-0.21 to 0.70]
Statistical Analysis 31: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.50 to 0.42]
Statistical Analysis 32: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.43 to 0.48]
Statistical Analysis 33: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 33]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.76, 95% CI 2-sided [0.26 to 1.26]
Statistical Analysis 34: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 33]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.21, 95% CI 2-sided [-0.29 to 0.70]
Statistical Analysis 35: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 33]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.55 to 0.44]
Statistical Analysis 36: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 33]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.43 to 0.56]
Statistical Analysis 37: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.89, 95% CI 2-sided [0.37 to 1.41]
Statistical Analysis 38: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.37, 95% CI 2-sided [-0.15 to 0.89]
Statistical Analysis 39: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.61 to 0.42]
Statistical Analysis 40: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.46 to 0.57]

24. Secondary Outcome: Change From Baseline in DAS28-4(CRP) at Week 12 (Descriptive Statistics)
Description: DAS28-4 (CRP) was calculated from the SJC and TJC using the 28 joints count and CRP (mg/L). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-3 (CRP) <= 3.2 implied low disease activity and >3.2 to 5.1 implied moderate to high disease activity, and DAS28-3 (CRP) <2.6 = remission.
Time Frame: Week 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | PF-04171327 1 mg | PF-04171327 5 mg | PF-04171327 10 mg | PF-04171327 15 mg | Prednisone 5 mg | Prednisone 10 mg | Placebo
Number analyzed (Participants) | 43 | 41 | 44 | 41 | 44 | 42 | 40
Units on a scale | -1.39 (1.31) | -1.56 (1.17) | -1.42 (1.19) | -1.38 (1.47) | -1.59 (1.22) | -1.80 (1.14) | -1.29 (1.21)

25. Secondary Outcome: Change From Baseline in SF-36v2 Mental Component Scores at Weeks 4 and 8 (Comparisons to Placebo, and Prednisone 10 mg)
Description: The 36 item Short Form Health Survey (SF-36) (Versions 2, acute version) is a 36 item generic health status measure. It measures 8 general health concepts: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. These concepts can also be summarized as physical component score (PCS) and mental component score (MCS). The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning). This questionnaire was completed by the participant prior to any procedures being performed at the visit, if possible. The form was then checked by site staff for completeness.
Time Frame: Weeks 4 and 8
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | PF-04171327 1 mg | PF-04171327 5 mg | PF-04171327 10 mg | PF-04171327 15 mg | Prednisone 5 mg | Prednisone 10 mg | Placebo
Number analyzed (Participants) | 45 | 47 | 45 | 48 | 45 | 46 | 47
Units on a scale
  Week 4: number analyzed (Participants) | 45 | 46 | 44 | 47 | 44 | 44 | 45
  Week 4 | 3.59 (1.28) | 4.53 (1.26) | 5.22 (1.30) | 5.74 (1.25) | 3.67 (1.29) | 7.23 (1.29) | 4.98 (1.28)
  Week 8: number analyzed (Participants) | 44 | 42 | 44 | 44 | 44 | 44 | 44
  Week 8 | 2.57 (1.39) | 6.07 (1.41) | 6.03 (1.40) | 6.47 (1.39) | 5.30 (1.40) | 8.76 (1.40) | 4.58 (1.39)
Statistical Analysis 1: Comparison: PF-04171327 1 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -1.38, 95% CI 2-sided [-4.94 to 2.17]
Statistical Analysis 2: Comparison: PF-04171327 5 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.45, 95% CI 2-sided [-3.98 to 3.08]
Statistical Analysis 3: Comparison: PF-04171327 10 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.24, 95% CI 2-sided [-3.34 to 3.82]
Statistical Analysis 4: Comparison: PF-04171327 15 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.76, 95% CI 2-sided [-2.75 to 4.28]
Statistical Analysis 5: Comparison: Prednisone 5 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = -1.31, 95% CI 2-sided [-4.88 to 2.27]
Statistical Analysis 6: Comparison: Prednisone 10 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = 2.25, 95% CI 2-sided [-1.32 to 5.82]
Statistical Analysis 7: Comparison: PF-04171327 1 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = -2.01, 95% CI 2-sided [-5.89 to 1.87]
Statistical Analysis 8: Comparison: PF-04171327 5 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = 1.49, 95% CI 2-sided [-2.41 to 5.40]
Statistical Analysis 9: Comparison: PF-04171327 10 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = 1.45, 95% CI 2-sided [-2.44 to 5.34]
Statistical Analysis 10: Comparison: PF-04171327 15 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = 1.89, 95% CI 2-sided [-1.98 to 5.76]
Statistical Analysis 11: Comparison: Prednisone 5 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.73, 95% CI 2-sided [-3.16 to 4.61]
Statistical Analysis 12: Comparison: Prednisone 10 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = 4.18, 95% CI 2-sided [0.29 to 8.06]
Statistical Analysis 13: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = -3.64, 95% CI 2-sided [-7.21 to -0.06]
Statistical Analysis 14: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = -2.70, 95% CI 2-sided [-6.25 to 0.85]
Statistical Analysis 15: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = -2.01, 95% CI 2-sided [-5.63 to 1.60]
Statistical Analysis 16: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = -1.49, 95% CI 2-sided [-5.02 to 2.05]
Statistical Analysis 17: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = -6.19, 95% CI 2-sided [-10.07 to -2.31]
Statistical Analysis 18: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = -2.69, 95% CI 2-sided [-6.60 to 1.23]
Statistical Analysis 19: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = -2.73, 95% CI 2-sided [-6.64 to 1.18]
Statistical Analysis 20: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = -2.29, 95% CI 2-sided [-6.16 to 1.58]

26. Secondary Outcome: Change From Baseline in SF-36v2 Mental Component Scores at Week 12 (Descriptive Statistics)
Description: as for outcome 25
Time Frame: Week 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | PF-04171327 1 mg | PF-04171327 5 mg | PF-04171327 10 mg | PF-04171327 15 mg | Prednisone 5 mg | Prednisone 10 mg | Placebo
Number analyzed (Participants) | 44 | 41 | 44 | 43 | 43 | 42 | 41
Units on a scale | 3.35 (11.99) | 4.19 (9.19) | 0.48 (8.97) | 2.72 (10.67) | 3.08 (12.91) | 6.11 (12.90) | 4.69 (10.72)

27. Secondary Outcome: Change From Baseline in SF-36v2 Physical Component Scores at Weeks 4 and 8 (Comparisons to Placebo, and Prednisone 10 mg)
Description: as for outcome 25
Time Frame: Weeks 4 and 8
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | PF-04171327 1 mg | PF-04171327 5 mg | PF-04171327 10 mg | PF-04171327 15 mg | Prednisone 5 mg | Prednisone 10 mg | Placebo
Number analyzed (Participants) | 45 | 47 | 45 | 48 | 45 | 46 | 47
Units on a scale
  Week 4: number analyzed (Participants) | 45 | 46 | 44 | 47 | 44 | 44 | 45
  Week 4 | 3.84 (0.92) | 5.00 (0.91) | 8.22 (0.93) | 6.83 (0.90) | 4.28 (0.93) | 7.51 (0.93) | 2.10 (0.92)
  Week 8: number analyzed (Participants) | 44 | 42 | 44 | 44 | 44 | 44 | 44
  Week 8 | 5.24 (1.03) | 7.85 (1.04) | 9.65 (1.03) | 7.15 (1.02) | 7.06 (1.03) | 9.62 (1.03) | 3.45 (1.03)
Statistical Analysis 1: Comparison: PF-04171327 1 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = 1.73, 95% CI 2-sided [-0.83 to 4.30]
Statistical Analysis 2: Comparison: PF-04171327 5 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = 2.90, 95% CI 2-sided [0.35 to 5.45]
Statistical Analysis 3: Comparison: PF-04171327 10 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = 6.12, 95% CI 2-sided [3.54 to 8.70]
Statistical Analysis 4: Comparison: PF-04171327 15 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = 4.73, 95% CI 2-sided [2.19 to 7.26]
Statistical Analysis 5: Comparison: Prednisone 5 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = 2.18, 95% CI 2-sided [-0.39 to 4.76]
Statistical Analysis 6: Comparison: Prednisone 10 mg vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Mean Difference (Final Values) = 5.41, 95% CI 2-sided [2.83 to 7.99]
Statistical Analysis 7: Comparison: PF-04171327 1 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = 1.79, 95% CI 2-sided [-1.08 to 4.65]
Statistical Analysis 8: Comparison: PF-04171327 5 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = 4.40, 95% CI 2-sided [1.52 to 7.28]
Statistical Analysis 9: Comparison: PF-04171327 10 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = 6.20, 95% CI 2-sided [3.33 to 9.07]
Statistical Analysis 10: Comparison: PF-04171327 15 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = 3.70, 95% CI 2-sided [0.85 to 6.55]
Statistical Analysis 11: Comparison: Prednisone 5 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = 3.61, 95% CI 2-sided [0.74 to 6.47]
Statistical Analysis 12: Comparison: Prednisone 10 mg vs Placebo; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; Mean Difference (Final Values) = 6.17, 95% CI 2-sided [3.29 to 9.04]
Statistical Analysis 13: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = -3.68, 95% CI 2-sided [-6.27 to -1.09]
Statistical Analysis 14: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = -2.51, 95% CI 2-sided [-5.07 to 0.05]
Statistical Analysis 15: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.71, 95% CI 2-sided [-1.88 to 3.30]
Statistical Analysis 16: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 29]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.68, 95% CI 2-sided [-3.23 to 1.87]
Statistical Analysis 17: Comparison: PF-04171327 1 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = -4.38, 95% CI 2-sided [-7.26 to -1.50]
Statistical Analysis 18: Comparison: PF-04171327 5 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = -1.76, 95% CI 2-sided [-4.65 to 1.12]
Statistical Analysis 19: Comparison: PF-04171327 10 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-2.84 to 2.91]
Statistical Analysis 20: Comparison: PF-04171327 15 mg vs Prednisone 10 mg; [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; Mean Difference (Final Values) = -2.47, 95% CI 2-sided [-5.33 to 0.39]

28. Secondary Outcome: Change From Baseline in SF-36v2 Physical Component Scores at Week 12 (Descriptive Statistics)
Description: as for outcome 25
Time Frame: Week 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | PF-04171327 1 mg | PF-04171327 5 mg | PF-04171327 10 mg | PF-04171327 15 mg | Prednisone 5 mg | Prednisone 10 mg | Placebo
Number analyzed (Participants) | 44 | 41 | 44 | 43 | 43 | 42 | 41
Units on a scale | 4.64 (8.21) | 5.39 (7.05) | 7.42 (8.56) | 3.91 (7.16) | 7.63 (7.95) | 5.85 (7.32) | 3.23 (4.80)

ADVERSE EVENTS:
Time Frame: 13 weeks
Description: All causality AEs and SAEs are included in this section. The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | PF-04171327 1 mg | PF-04171327 5 mg | PF-04171327 10 mg | PF-04171327 15 mg | Prednisone 5 mg | Prednisone 10 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/45 | 1/47 | 2/45 | 2/48 | 0/45 | 2/46 | 2/47
Other Adverse Events (participants affected / at risk) | 20/45 | 18/47 | 22/45 | 16/48 | 16/45 | 19/46 | 16/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04171327 1 mg (N=45) | PF-04171327 5 mg (N=47) | PF-04171327 10 mg (N=45) | PF-04171327 15 mg (N=48) | Prednisone 5 mg (N=45) | Prednisone 10 mg (N=46) | Placebo (N=47)
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04171327 1 mg (N=45) | PF-04171327 5 mg (N=47) | PF-04171327 10 mg (N=45) | PF-04171327 15 mg (N=48) | Prednisone 5 mg (N=45) | Prednisone 10 mg (N=46) | Placebo (N=47)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Monocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Goitre (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Astigmatism (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Presbyopia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 2 | 2 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1
Oral discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 1 | 0 | 1 | 1 | 0 | 2 | 0
Drug ineffective (General disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 1
Face oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Local swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abscess bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 0 | 1
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 3 | 3 | 2 | 0 | 1 | 1
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 1
Pharyngitis bacterial (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 3 | 2 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Viral rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1 | 4 | 0 | 0 | 3 | 3
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 1 | 0 | 0 | 2 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Blood creatinine decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 1 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 1 | 5 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 1 | 0 | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 3 | 0 | 1
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 4 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Microalbuminuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Polymenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Knee operation (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 3 | 0 | 1 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0
Varicose vein (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.